CLINICAL TRIAL: NCT05415410
Title: A Randomized, Single-blind Trial to Evaluate the Safety and Efficacy of Apraglutide in Subjects With Grade II to IV (MAGIC) Steroid Refractory Gastrointestinal (GI) Acute Graft Versus Host Disease on Best Available Therapy
Brief Title: Proof-of-concept Trial of Apraglutide in Acute Graft Versus Host Disease (aGVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TA799-101
Record Dates: First submitted 2022-02-08; First posted 2022-06-13 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: GVHD
Keywords: Graft versus host disease; GVHD; GVHD, Acute; Steroid-refractory aGVHD; Gastrointestinal-GVHD; GI-GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — apraglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Apraglutide Low Dose (Experimental): Low-dose, weight-based apraglutide subcutaneous (SC) injections (1.4 to 3.5 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight of more than 50.0 kg.
  Interventions: Drug: Apraglutide
- Apraglutide High Dose (Experimental): High-dose, weight-based apraglutide SC injections (3.5 to 7.6 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight of more than 50.0 kg.
  Interventions: Drug: Apraglutide
- Apraglutide Standard Dose (Experimental): Standard-dose apraglutide SC injections (1.4 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight between 40.0 kg to 49.9 kg.
  Interventions: Drug: Apraglutide

INTERVENTIONS:
Drug: Apraglutide — Apraglutide is a new, synthetic glucagon-like peptide 2 (GLP-2) receptor agonist which acts as a gut targeted regenerative approach that is intestinotrophic with a mode of action that improves absorption and enhances gut barrier function.

SUMMARY:
The aim of this trial is to assess safety and efficacy of apraglutide in subjects with steroid refractory gastrointestinal aGVHD.

DETAILED DESCRIPTION:
This is an international, multicenter, randomized proof-of-concept trial to evaluate safety, tolerability, efficacy, durability of response, and clinical outcomes of apraglutide administration to subjects with steroid-refractory (SR) aGVHD of the lower GI tract being treated with systemic steroids (SS) and ruxolitinib (RUX).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent and agree to follow the details of participation as outlined in the protocol
* Male or female subjects aged 12 years or above at the time of consent and who weigh a minimum of 40 kg. Only subjects aged 18 years and above will be included in Germany.
* Clinically confirmed steroid refractory lower GI-aGVHD (MAGIC stage 1-4) prior to randomization
* Have undergone alloSCT from any donor source, any conditioning regimen
* Treated with SS plus RUX (RUX starts concomitantly to apraglutide or a maximum of 72 hours before apraglutide initiation)
* Women of childbearing potential (WOCBP): highly effective method of contraception and refrain from donating eggs during the trial and for 4 weeks after the End of Trial (EOT) visit
* Male subjects with partner WOCBP: contraception and abstention from sperm donation during the trial and for 2 weeks after the EOT visit

Exclusion Criteria:

* Treatment with any systemic GVHD therapy other than SS and RUX including methotrexate and mycophenolate mofetil at the time of randomization / Day 0
* Concomitant treatment with Janus kinase inhibitor other than RUX at the time of randomization
* Failed alloSCT due to relapse of underlying malignant disease
* Presence of SR GI-aGVHD occurring after donor lymphocyte infusion for pre-emptive treatment of malignancy recurrence
* Any use of enteral glutamine or GLP analogs or known ADA, within 6 months prior to randomization / Day 0
* Significant organ system failures (respiratory renal hepatic and cardiac)
* Presence of relapsed primary malignancy or treatment for relapse after alloHSCT
* Presence or history of GI tumors (including the hepatobiliary system and pancreas) within the last five years before randomization
* Presence of colonic polyps not removed
* Active clinically uncontrolled infection or active tuberculosis
* Known chronic GVHD
* Known active GI inflammation not related to GI-aGVHD
* Major abdominal surgery in the last 6-months prior to randomization or history of clinically significant intestinal adhesions
* Abnormal liver function tests

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (13):
- United States (5):
  - Stanford Cancer Center, Stanford, California
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
  - South Austin Medical Center, Austin, Texas
- Germany (6):
  - Universitätsklinikum Köln (AoeR), Cologne
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Martin Luther Universität Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsmedizin der Johannes Gutenberg - Universität Mainz, Mainz
- Instituto Portugues de Oncologia do Porto Francisco Gentil, Porto, Portugal
- Hospital Universitario Virgen del Rocio, Seville, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Started | 15 | 15 | 1
Completed | 2 | 1 | 0
Not Completed | 13 | 14 | 1
Not completed — Death | 3 | 6 | 1
Not completed — Trial Terminated by Sponsor | 1 | 5 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Physician Decision due to Non-Compliance | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Pregnancy | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Apraglutide Low Dose: Low-dose, weight-based apraglutide SC injections (1.4 to 3.5 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight of more than 50.0 kg.
- Total: Total of all reporting groups
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose | Total
Number analyzed (Participants) | 15 | 15 | 1 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.00) | 62.0 (9.68) | 52.0 (NA) — 1 participant in this group. | 60.2 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 1 | 12
  Male | 11 | 8 | 0 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 1 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 14 | 1 | 29
  Asian | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE=any untoward medical occurrence which does not necessarily have a causal relationship with study drug. Serious AE (SAE)=any AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a neonate/infant born to a mother or father exposed to study drug; is a clinically significant event in the Investigator's judgment. Treatment-emergent AE (TEAE)=AE with a start on or after the first administration of apraglutide (or present prior to the first dose of apraglutide but worsening in severity after starting treatment relative to the pre-treatment state) up to 28 days after the last dose of apraglutide. Pre-treatment AE=occurs after informed consent and before first dose; post-treatment AE=occurs after 28 days from last dose. AE are graded as follows: mild (1), moderate (2), severe (3), life-threatening (4), death (5).
Time Frame: Screening (up to 12 weeks) through End of Trial (up to 2 years/104 weeks) for a total of up to 116 weeks
Population: Safety Analysis Set: All the randomized participants exposed to at least 1 dose of apraglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Any Pre-Treatment AEs | 5 | 8 | 0
  Any Pre-Treatment AEs: Grade 1 | 0 | 1 | 0
  Any Pre-Treatment AEs: Grade 2 | 1 | 2 | 0
  Any Pre-Treatment AEs: Grade 3 | 4 | 4 | 0
  Any Pre-Treatment AEs: Grade 4 | 0 | 1 | 0
  Any Pre-Treatment AEs: Grade 5 | 0 | 0 | 0
  Any Pre-Treatment AEs: >= Grade 3 | 4 | 5 | 0
  Any Pre-Treatment AE Leading to Death | 0 | 0 | 0
  Any Serious Pre-Treatment AEs | 0 | 1 | 0
  Any TEAEs | 15 | 15 | 1
  Any TEAEs Grade 1 | 0 | 0 | 0
  Any TEAEs Grade 2 | 2 | 0 | 0
  Any TEAEs Grade 3 | 10 | 4 | 0
  Any TEAEs Grade 4 | 1 | 5 | 0
  Any TEAEs Grade 5 | 2 | 6 | 1
  Any TEAEs >= Grade 3 | 13 | 15 | 1
  Any TEAE Leading to Death | 2 | 6 | 1
  Any Drug-Related TEAEs | 5 | 4 | 0
  Any Drug-Related TEAEs Grade 1 | 0 | 1 | 0
  Any Drug-Related TEAEs Grade 2 | 2 | 0 | 0
  Any Drug-Related TEAEs Grade 3 | 3 | 2 | 0
  Any Drug-Related TEAEs Grade 4 | 0 | 1 | 0
  Any Drug-Related TEAEs Grade 5 | 0 | 0 | 0
  Any Drug-Related TEAEs >= Grade 3 | 3 | 3 | 0
  Any Serious TEAEs | 6 | 15 | 1
  Any Drug-Related Serious TEAEs | 1 | 0 | 0
  Any TEAEs Leading to Dose Reduction | 0 | 0 | 0
  Any TEAEs Leading to Dose Interruption | 3 | 4 | 0
  Any TEAEs Leading to Permanent Discontinuation of Apraglutide | 5 | 6 | 1
  Any TEAEs Meeting Trial Stopping Criteria | 5 | 0 | 0
  Any TEAEs Leading to Discontinuation from Trial | 3 | 6 | 1
  Any Post-Treatment AEs | 10 | 8 | 1
  Any Post-Treatment AEs Grade 1 | 0 | 1 | 0
  Any Post-Treatment AEs Grade 2 | 4 | 1 | 0
  Any Post-Treatment AEs Grade 3 | 3 | 5 | 1
  Any Post-Treatment AEs Grade 4 | 2 | 0 | 0
  Any Post-Treatment AEs Grade 5 | 1 | 1 | 0
  Any Post-Treatment AEs >= Grade 3 | 6 | 6 | 1
  Any Post-Treatment AEs Leading to Death | 1 | 1 | 0
  Any Drug-Related Post-Treatment AEs | 0 | 2 | 0
  Any Drug-Related Post-Treatment AEs Grade 1 | 0 | 0 | 0
  Any Drug-Related Post-Treatment AEs Grade 2 | 0 | 2 | 0
  Any Drug-Related Post-Treatment AEs Grade 3 | 0 | 0 | 0
  Any Drug-Related Post-Treatment AEs Grade 4 | 0 | 0 | 0
  Any Drug-Related Post-Treatment AEs Grade 5 | 0 | 0 | 0
  Any Drug-Related Post-Treatment AEs >= Grade 3 | 0 | 0 | 0
  Any Serious Post-Treatment AEs | 6 | 2 | 0
  Any Drug-Related Serious Post-Treatment AEs | 0 | 0 | 0
  Any Post-Treatment AEs Meeting Trial Stopping Criteria | 0 | 0 | 0
  Any Post-Treatment AEs Leading to Discontinuation From Trial | 2 | 1 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) is an AE of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring, additional information, and rapid communication by the Investigator to the Sponsor is appropriate. AESIs include:
  * Injection site reactions
  * Gastrointestinal obstructions
  * Gallbladder, biliary, and pancreatic disease
  * Fluid overload
  * Colorectal polyps
  * Newly diagnosed malignancies
  * Systemic hypersensitivity
Time Frame: From first dose of study drug through End of Trial (up to 2 years/104 weeks) for a total of up to 116 weeks
Population: Safety Analysis Set: All the randomized participants exposed to at least 1 dose of apraglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Gastrointestinal Obstructions | 3 | 4 | 0
  Fluid Overload | 2 | 2 | 0
  Gall Bladder, Biliary and Pancreatic Disease | 0 | 1 | 0
  Colorectal Polyps | 0 | 0 | 0
  Injection Site Reactions | 0 | 0 | 0
  Newly Diagnosed Malignancy | 0 | 0 | 0
  Systemic Hypersensitivity | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline Over Time in Vital Signs
Description: Systolic Blood Pressure:
  * High is defined as >= 160 mmHg AND >=20 mmHg increase from baseline
  * Low is defined as <= 90 mmHg AND >=20 mmHg decrease from baseline
  Diastolic Blood Pressure:
  * High is defined as >= 100 mmHg AND >=15 mmHg increase from baseline
  * Low is defined as <= 50 mmHg AND >=15 mmHg decrease from baseline
  Heart Rate:
  * High is defined as >= 120 bpm AND >= 15 bpm increase from baseline
  * Low is defined as <= 50 bpm AND >= 15 bpm decrease from baseline
  Baseline is defined as the last measurement prior to the first dose of apraglutide. Minimum post-baseline is defined as the minimum measurement after the first dose of apraglutide. Maximum post-baseline is defined as the maximum measurement after the first dose of apraglutide.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 13, 17, 21, 26, 52, End of Treatment (up to Week 25), Week 104/End of Trial
Population: Safety Analysis Set: All the randomized participants exposed to at least 1 dose of apraglutide. Participants with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Systolic Blood Pressure Week 1 : High | 0 | 0 | 0
  Systolic Blood Pressure Week 1 : Low | 0 | 0 | 0
  Systolic Blood Pressure Week 1 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 2 : High: number analyzed (Participants) | 14 | 14 | 1
  Systolic Blood Pressure Week 2 : High | 1 | 0 | 0
  Systolic Blood Pressure Week 2 : Low: number analyzed (Participants) | 14 | 14 | 1
  Systolic Blood Pressure Week 2 : Low | 0 | 1 | 0
  Systolic Blood Pressure Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  Systolic Blood Pressure Week 2 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 3 : High: number analyzed (Participants) | 13 | 13 | 1
  Systolic Blood Pressure Week 3 : High | 0 | 2 | 0
  Systolic Blood Pressure Week 3 : Low: number analyzed (Participants) | 13 | 13 | 1
  Systolic Blood Pressure Week 3 : Low | 1 | 0 | 0
  Systolic Blood Pressure Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  Systolic Blood Pressure Week 3 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 4 : High: number analyzed (Participants) | 12 | 12 | 1
  Systolic Blood Pressure Week 4 : High | 0 | 0 | 0
  Systolic Blood Pressure Week 4 : Low: number analyzed (Participants) | 12 | 12 | 1
  Systolic Blood Pressure Week 4 : Low | 0 | 0 | 0
  Systolic Blood Pressure Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  Systolic Blood Pressure Week 4 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 6 : High: number analyzed (Participants) | 11 | 9 | 1
  Systolic Blood Pressure Week 6 : High | 0 | 0 | 0
  Systolic Blood Pressure Week 6 : Low: number analyzed (Participants) | 11 | 9 | 1
  Systolic Blood Pressure Week 6 : Low | 0 | 0 | 0
  Systolic Blood Pressure Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  Systolic Blood Pressure Week 6 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 8 : High: number analyzed (Participants) | 10 | 8 | 1
  Systolic Blood Pressure Week 8 : High | 0 | 0 | 0
  Systolic Blood Pressure Week 8 : Low: number analyzed (Participants) | 10 | 8 | 1
  Systolic Blood Pressure Week 8 : Low | 0 | 1 | 0
  Systolic Blood Pressure Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  Systolic Blood Pressure Week 8 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 13 : High: number analyzed (Participants) | 8 | 8 | 1
  Systolic Blood Pressure Week 13 : High | 0 | 0 | 0
  Systolic Blood Pressure Week 13 : Low: number analyzed (Participants) | 8 | 8 | 1
  Systolic Blood Pressure Week 13 : Low | 0 | 0 | 0
  Systolic Blood Pressure Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  Systolic Blood Pressure Week 13 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 17 : High: number analyzed (Participants) | 7 | 7 | 1
  Systolic Blood Pressure Week 17 : High | 0 | 0 | 0
  Systolic Blood Pressure Week 17 : Low: number analyzed (Participants) | 7 | 7 | 1
  Systolic Blood Pressure Week 17 : Low | 0 | 0 | 0
  Systolic Blood Pressure Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  Systolic Blood Pressure Week 17 : Missing | 0 | 0 | 0
  Systolic Blood Pressure Week 21 : High: number analyzed (Participants) | 4 | 7 | 0
  Systolic Blood Pressure Week 21 : High | 0 | 0 |
  Systolic Blood Pressure Week 21 : Low: number analyzed (Participants) | 4 | 7 | 0
  Systolic Blood Pressure Week 21 : Low | 0 | 0 |
  Systolic Blood Pressure Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  Systolic Blood Pressure Week 21 : Missing | 0 | 0 |
  Systolic Blood Pressure Week 26 : High: number analyzed (Participants) | 4 | 5 | 0
  Systolic Blood Pressure Week 26 : High | 0 | 0 |
  Systolic Blood Pressure Week 26 : Low: number analyzed (Participants) | 4 | 5 | 0
  Systolic Blood Pressure Week 26 : Low | 0 | 0 |
  Systolic Blood Pressure Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  Systolic Blood Pressure Week 26 : Missing | 0 | 0 |
  Systolic Blood Pressure Week 52 : High: number analyzed (Participants) | 2 | 0 | 0
  Systolic Blood Pressure Week 52 : High | 0 |  |
  Systolic Blood Pressure Week 52 : Low: number analyzed (Participants) | 2 | 0 | 0
  Systolic Blood Pressure Week 52 : Low | 0 |  |
  Systolic Blood Pressure Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  Systolic Blood Pressure Week 52 : Missing | 0 |  |
  Systolic Blood Pressure End of Treatment : High: number analyzed (Participants) | 0 | 2 | 0
  Systolic Blood Pressure End of Treatment : High |  | 1 |
  Systolic Blood Pressure End of Treatment : Low: number analyzed (Participants) | 0 | 2 | 0
  Systolic Blood Pressure End of Treatment : Low |  | 0 |
  Systolic Blood Pressure End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  Systolic Blood Pressure End of Treatment : Missing |  | 0 |
  Systolic Blood Pressure Week 104/End of Trial : High: number analyzed (Participants) | 5 | 1 | 0
  Systolic Blood Pressure Week 104/End of Trial : High | 0 | 0 |
  Systolic Blood Pressure Week 104/End of Trial : Low: number analyzed (Participants) | 5 | 1 | 0
  Systolic Blood Pressure Week 104/End of Trial : Low | 1 | 0 |
  Systolic Blood Pressure Week 104/End of Trial : Missing: number analyzed (Participants) | 5 | 1 | 0
  Systolic Blood Pressure Week 104/End of Trial : Missing | 0 | 0 |
  Systolic Blood Pressure Minimum Post-Baseline Value : High | 0 | 0 | 0
  Systolic Blood Pressure Minimum Post-Baseline Value : Low | 3 | 1 | 0
  Systolic Blood Pressure Minimum Post-Baseline Value : Missing | 0 | 0 | 0
  Systolic Blood Pressure Maximum Post-Baseline Value : High | 1 | 2 | 0
  Systolic Blood Pressure Maximum Post-Baseline Value : Low | 0 | 0 | 0
  Systolic Blood Pressure Maximum Post-Baseline Value : Missing | 0 | 0 | 0
  Systolic Blood Pressure Last Post-Baseline Value : High | 0 | 1 | 0
  Systolic Blood Pressure Last Post-Baseline Value : Low | 1 | 0 | 0
  Systolic Blood Pressure Last Post-Baseline Value : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 1 : High | 0 | 0 | 0
  Diastolic Blood Pressure Week 1 : Low | 1 | 0 | 0
  Diastolic Blood Pressure Week 1 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 2 : High: number analyzed (Participants) | 14 | 14 | 1
  Diastolic Blood Pressure Week 2 : High | 0 | 0 | 0
  Diastolic Blood Pressure Week 2 : Low: number analyzed (Participants) | 14 | 14 | 1
  Diastolic Blood Pressure Week 2 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  Diastolic Blood Pressure Week 2 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 3 : High: number analyzed (Participants) | 13 | 13 | 1
  Diastolic Blood Pressure Week 3 : High | 0 | 1 | 0
  Diastolic Blood Pressure Week 3 : Low: number analyzed (Participants) | 13 | 13 | 1
  Diastolic Blood Pressure Week 3 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  Diastolic Blood Pressure Week 3 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 4 : High: number analyzed (Participants) | 12 | 12 | 1
  Diastolic Blood Pressure Week 4 : High | 0 | 1 | 0
  Diastolic Blood Pressure Week 4 : Low: number analyzed (Participants) | 12 | 12 | 1
  Diastolic Blood Pressure Week 4 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  Diastolic Blood Pressure Week 4 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 6 : High: number analyzed (Participants) | 11 | 9 | 1
  Diastolic Blood Pressure Week 6 : High | 0 | 0 | 0
  Diastolic Blood Pressure Week 6 : Low: number analyzed (Participants) | 11 | 9 | 1
  Diastolic Blood Pressure Week 6 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  Diastolic Blood Pressure Week 6 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 8 : High: number analyzed (Participants) | 10 | 8 | 1
  Diastolic Blood Pressure Week 8 : High | 0 | 0 | 0
  Diastolic Blood Pressure Week 8 : Low: number analyzed (Participants) | 10 | 8 | 1
  Diastolic Blood Pressure Week 8 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  Diastolic Blood Pressure Week 8 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 13 : High: number analyzed (Participants) | 8 | 8 | 1
  Diastolic Blood Pressure Week 13 : High | 0 | 0 | 0
  Diastolic Blood Pressure Week 13 : Low: number analyzed (Participants) | 8 | 8 | 1
  Diastolic Blood Pressure Week 13 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  Diastolic Blood Pressure Week 13 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 17 : High: number analyzed (Participants) | 7 | 7 | 1
  Diastolic Blood Pressure Week 17 : High | 0 | 0 | 0
  Diastolic Blood Pressure Week 17 : Low: number analyzed (Participants) | 7 | 7 | 1
  Diastolic Blood Pressure Week 17 : Low | 0 | 0 | 0
  Diastolic Blood Pressure Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  Diastolic Blood Pressure Week 17 : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Week 21 : High: number analyzed (Participants) | 4 | 7 | 0
  Diastolic Blood Pressure Week 21 : High | 0 | 0 |
  Diastolic Blood Pressure Week 21 : Low: number analyzed (Participants) | 4 | 7 | 0
  Diastolic Blood Pressure Week 21 : Low | 0 | 0 |
  Diastolic Blood Pressure Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  Diastolic Blood Pressure Week 21 : Missing | 0 | 0 |
  Diastolic Blood Pressure Week 26 : High: number analyzed (Participants) | 4 | 5 | 0
  Diastolic Blood Pressure Week 26 : High | 0 | 0 |
  Diastolic Blood Pressure Week 26 : Low: number analyzed (Participants) | 4 | 5 | 0
  Diastolic Blood Pressure Week 26 : Low | 0 | 0 |
  Diastolic Blood Pressure Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  Diastolic Blood Pressure Week 26 : Missing | 0 | 0 |
  Diastolic Blood Pressure Week 52 : High: number analyzed (Participants) | 2 | 0 | 0
  Diastolic Blood Pressure Week 52 : High | 0 |  |
  Diastolic Blood Pressure Week 52 : Low: number analyzed (Participants) | 2 | 0 | 0
  Diastolic Blood Pressure Week 52 : Low | 0 |  |
  Diastolic Blood Pressure Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  Diastolic Blood Pressure Week 52 : Missing | 0 |  |
  Diastolic Blood Pressure End of Treatment : High: number analyzed (Participants) | 0 | 2 | 0
  Diastolic Blood Pressure End of Treatment : High |  | 0 |
  Diastolic Blood Pressure End of Treatment : Low: number analyzed (Participants) | 0 | 2 | 0
  Diastolic Blood Pressure End of Treatment : Low |  | 0 |
  Diastolic Blood Pressure End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  Diastolic Blood Pressure End of Treatment : Missing |  | 0 |
  Diastolic Blood Pressure Week 104 : High: number analyzed (Participants) | 5 | 1 | 0
  Diastolic Blood Pressure Week 104 : High | 0 | 0 |
  Diastolic Blood Pressure Week 104 : Low: number analyzed (Participants) | 5 | 1 | 0
  Diastolic Blood Pressure Week 104 : Low | 0 | 0 |
  Diastolic Blood Pressure Week 104 : Missing: number analyzed (Participants) | 5 | 1 | 0
  Diastolic Blood Pressure Week 104 : Missing | 0 | 0 |
  Diastolic Blood Pressure Minimum Post-Baseline Value : High | 0 | 0 | 0
  Diastolic Blood Pressure Minimum Post-Baseline Value : Low | 1 | 0 | 0
  Diastolic Blood Pressure Minimum Post-Baseline Value : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Maximum Post-Baseline Value : High | 0 | 1 | 0
  Diastolic Blood Pressure Maximum Post-Baseline Value : Low | 0 | 0 | 0
  Diastolic Blood Pressure Maximum Post-Baseline Value : Missing | 0 | 0 | 0
  Diastolic Blood Pressure Last Post-Baseline Value : High | 0 | 0 | 0
  Diastolic Blood Pressure Last Post-Baseline Value : Low | 0 | 0 | 0
  Diastolic Blood Pressure Last Post-Baseline Value : Missing | 0 | 0 | 0
  Heart Rate Week 1 : High | 0 | 0 | 0
  Heart Rate Week 1 : Low | 0 | 0 | 0
  Heart Rate Week 1 : Missing | 0 | 0 | 0
  Heart Rate Week 2 : High: number analyzed (Participants) | 14 | 14 | 1
  Heart Rate Week 2 : High | 0 | 0 | 0
  Heart Rate Week 2 : Low: number analyzed (Participants) | 14 | 14 | 1
  Heart Rate Week 2 : Low | 0 | 0 | 0
  Heart Rate Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  Heart Rate Week 2 : Missing | 0 | 0 | 0
  Heart Rate Week 3 : High: number analyzed (Participants) | 13 | 13 | 1
  Heart Rate Week 3 : High | 2 | 1 | 0
  Heart Rate Week 3 : Low: number analyzed (Participants) | 13 | 13 | 1
  Heart Rate Week 3 : Low | 0 | 0 | 0
  Heart Rate Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  Heart Rate Week 3 : Missing | 0 | 0 | 0
  Heart Rate Week 4 : High: number analyzed (Participants) | 12 | 12 | 1
  Heart Rate Week 4 : High | 0 | 0 | 0
  Heart Rate Week 4 : Low: number analyzed (Participants) | 12 | 12 | 1
  Heart Rate Week 4 : Low | 0 | 0 | 0
  Heart Rate Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  Heart Rate Week 4 : Missing | 0 | 0 | 0
  Heart Rate Week 6 : High: number analyzed (Participants) | 11 | 9 | 1
  Heart Rate Week 6 : High | 0 | 0 | 0
  Heart Rate Week 6 : Low: number analyzed (Participants) | 11 | 9 | 1
  Heart Rate Week 6 : Low | 0 | 0 | 0
  Heart Rate Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  Heart Rate Week 6 : Missing | 0 | 0 | 0
  Heart Rate Week 8 : High: number analyzed (Participants) | 10 | 8 | 1
  Heart Rate Week 8 : High | 0 | 0 | 0
  Heart Rate Week 8 : Low: number analyzed (Participants) | 10 | 8 | 1
  Heart Rate Week 8 : Low | 0 | 0 | 0
  Heart Rate Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  Heart Rate Week 8 : Missing | 0 | 0 | 0
  Heart Rate Week 13 : High: number analyzed (Participants) | 8 | 8 | 1
  Heart Rate Week 13 : High | 0 | 0 | 0
  Heart Rate Week 13 : Low: number analyzed (Participants) | 8 | 8 | 1
  Heart Rate Week 13 : Low | 0 | 0 | 0
  Heart Rate Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  Heart Rate Week 13 : Missing | 0 | 0 | 0
  Heart Rate Week 17 : High: number analyzed (Participants) | 7 | 7 | 1
  Heart Rate Week 17 : High | 0 | 0 | 0
  Heart Rate Week 17 : Low: number analyzed (Participants) | 7 | 7 | 1
  Heart Rate Week 17 : Low | 0 | 0 | 0
  Heart Rate Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  Heart Rate Week 17 : Missing | 1 | 0 | 0
  Heart Rate Week 21 : High: number analyzed (Participants) | 4 | 7 | 0
  Heart Rate Week 21 : High | 0 | 0 |
  Heart Rate Week 21 : Low: number analyzed (Participants) | 4 | 7 | 0
  Heart Rate Week 21 : Low | 0 | 1 |
  Heart Rate Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  Heart Rate Week 21 : Missing | 0 | 0 |
  Heart Rate Week 26 : High: number analyzed (Participants) | 4 | 5 | 0
  Heart Rate Week 26 : High | 0 | 0 |
  Heart Rate Week 26 : Low: number analyzed (Participants) | 4 | 5 | 0
  Heart Rate Week 26 : Low | 0 | 0 |
  Heart Rate Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  Heart Rate Week 26 : Missing | 0 | 0 |
  Heart Rate Week 52 : High: number analyzed (Participants) | 2 | 0 | 0
  Heart Rate Week 52 : High | 0 |  |
  Heart Rate Week 52 : Low: number analyzed (Participants) | 2 | 0 | 0
  Heart Rate Week 52 : Low | 0 |  |
  Heart Rate Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  Heart Rate Week 52 : Missing | 0 |  |
  Heart Rate End of Treatment : High: number analyzed (Participants) | 0 | 2 | 0
  Heart Rate End of Treatment : High |  | 0 |
  Heart Rate End of Treatment : Low: number analyzed (Participants) | 0 | 2 | 0
  Heart Rate End of Treatment : Low |  | 0 |
  Heart Rate End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  Heart Rate End of Treatment : Missing |  | 0 |
  Heart Rate Week 104/End of Trial : High: number analyzed (Participants) | 5 | 1 | 0
  Heart Rate Week 104/End of Trial : High | 0 | 0 |
  Heart Rate Week 104/End of Trial : Low: number analyzed (Participants) | 5 | 1 | 0
  Heart Rate Week 104/End of Trial : Low | 0 | 0 |
  Heart Rate Week 104/End of Trial : Missing: number analyzed (Participants) | 5 | 1 | 0
  Heart Rate Week 104/End of Trial : Missing | 0 | 0 |
  Heart Rate Minimum Post-Baseline Value : High | 0 | 0 | 0
  Heart Rate Minimum Post-Baseline Value : Low | 0 | 1 | 0
  Heart Rate Minimum Post-Baseline Value : Missing | 0 | 0 | 0
  Heart Rate Maximum Post-Baseline Value : High | 2 | 1 | 0
  Heart Rate Maximum Post-Baseline Value : Low | 0 | 0 | 0
  Heart Rate Maximum Post-Baseline Value : Missing | 0 | 0 | 0
  Heart Rate Last Post-Baseline Value : High | 1 | 0 | 0
  Heart Rate Last Post-Baseline Value : Low | 0 | 0 | 0
  Heart Rate Last Post-Baseline Value : Missing | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline Over Time in QT Corrected for Heart Rate Using Fridericia's Formula (QTcF)
Description: Baseline is defined as the last measurement prior to the first dose of apraglutide. Minimum post-baseline is defined as the minimum measurement after the first dose of apraglutide. Maximum post-baseline is defined as the maximum measurement after the first dose of apraglutide.
Time Frame: Baseline, Weeks 26, 52, 104/End of Trial
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 14 | 13 | 1
Participants
  Baseline : QTcF Interval > 450 - 480 msec | 2 | 2 | 0
  Baseline : QTcF Interval > 480 - 500 msec | 0 | 1 | 0
  Baseline : QTcF Interval > 500 msec | 0 | 0 | 0
  Baseline : Increase from Baseline QTcF Interval > 30 - 60 msec | 0 | 0 | 0
  Baseline : Increase from Baseline QTcF Interval > 60 msec | 0 | 0 | 0
  Baseline : Missing | 0 | 0 | 0
  Week 26 : QTcF Interval > 450 - 480 msec: number analyzed (Participants) | 3 | 3 | 0
  Week 26 : QTcF Interval > 450 - 480 msec | 0 | 0 |
  Week 26 : QTcF Interval > 480 - 500 msec: number analyzed (Participants) | 3 | 3 | 0
  Week 26 : QTcF Interval > 480 - 500 msec | 0 | 0 |
  Week 26 : QTcF Interval > 500 msec: number analyzed (Participants) | 3 | 3 | 0
  Week 26 : QTcF Interval > 500 msec | 0 | 0 |
  Week 26 : Increase from Baseline QTcF Interval > 30 - 60 msec: number analyzed (Participants) | 3 | 13 | 0
  Week 26 : Increase from Baseline QTcF Interval > 30 - 60 msec | 0 | 0 |
  Week 26 : Increase from Baseline QTcF Interval > 60 msec: number analyzed (Participants) | 3 | 13 | 0
  Week 26 : Increase from Baseline QTcF Interval > 60 msec | 0 | 0 |
  Week 26 : Missing: number analyzed (Participants) | 3 | 13 | 0
  Week 26 : Missing | 0 | 0 |
  Week 52 : QTcF Interval > 450 - 480 msec: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : QTcF Interval > 450 - 480 msec | 0 |  |
  Week 52 : QTcF Interval > 480 - 500 msec: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : QTcF Interval > 480 - 500 msec | 0 |  |
  Week 52 : QTcF Interval > 500 msec: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : QTcF Interval > 500 msec | 0 |  |
  Week 52 : Increase from Baseline QTcF Interval > 30 - 60 msec: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : Increase from Baseline QTcF Interval > 30 - 60 msec | 1 |  |
  Week 52 : Increase from Baseline QTcF Interval > 60 msec: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : Increase from Baseline QTcF Interval > 60 msec | 0 |  |
  Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : Missing | 0 |  |
  Week 104/End of Trial : QTcF Interval > 450 - 480 msec: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : QTcF Interval > 450 - 480 msec | 0 | 0 |
  Week 104/End of Trial : QTcF Interval > 480 - 500 msec: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : QTcF Interval > 480 - 500 msec | 0 | 0 |
  Week 104/End of Trial : QTcF Interval > 500 msec: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : QTcF Interval > 500 msec | 0 | 0 |
  Week 104/End of Trial : Increase from Baseline QTcF Interval > 30 - 60 msec: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Increase from Baseline QTcF Interval > 30 - 60 msec | 0 | 0 |
  Week 104/End of Trial : Increase from Baseline QTcF Interval > 60 msec: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Increase from Baseline QTcF Interval > 60 msec | 0 | 0 |
  Week 104/End of Trial : Missing: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Missing | 0 | 1 |
  Minimum Post-Baseline Value : QTcF Interval > 450 - 480 msec: number analyzed (Participants) | 7 | 5 | 0
  Minimum Post-Baseline Value : QTcF Interval > 450 - 480 msec | 0 | 0 |
  Minimum Post-Baseline Value : QTcF Interval > 480 - 500 msec: number analyzed (Participants) | 7 | 5 | 0
  Minimum Post-Baseline Value : QTcF Interval > 480 - 500 msec | 0 | 0 |
  Minimum Post-Baseline Value : QTcF Interval > 500 msec: number analyzed (Participants) | 7 | 5 | 0
  Minimum Post-Baseline Value : QTcF Interval > 500 msec | 0 | 0 |
  Minimum Post-Baseline Value : Increase from Baseline QTcF Interval > 30 - 60 msec: number analyzed (Participants) | 7 | 5 | 0
  Minimum Post-Baseline Value : Increase from Baseline QTcF Interval > 30 - 60 msec | 0 | 0 |
  Minimum Post-Baseline Value : Increase from Baseline QTcF Interval > 60 msec: number analyzed (Participants) | 7 | 5 | 0
  Minimum Post-Baseline Value : Increase from Baseline QTcF Interval > 60 msec | 0 | 0 |
  Minimum Post-Baseline Value : Missing: number analyzed (Participants) | 7 | 5 | 0
  Minimum Post-Baseline Value : Missing | 0 | 1 |
  Maximum Post-Baseline Value : QTcF Interval > 450 - 480 msec: number analyzed (Participants) | 7 | 5 | 0
  Maximum Post-Baseline Value : QTcF Interval > 450 - 480 msec | 0 | 0 |
  Maximum Post-Baseline Value : QTcF Interval > 480 - 500 msec: number analyzed (Participants) | 7 | 5 | 0
  Maximum Post-Baseline Value : QTcF Interval > 480 - 500 msec | 0 | 0 |
  Maximum Post-Baseline Value : QTcF Interval > 500 msec: number analyzed (Participants) | 7 | 5 | 0
  Maximum Post-Baseline Value : QTcF Interval > 500 msec | 0 | 0 |
  Maximum Post-Baseline Value : Increase from Baseline QTcF Interval > 30 - 60 msec: number analyzed (Participants) | 7 | 5 | 0
  Maximum Post-Baseline Value : Increase from Baseline QTcF Interval > 30 - 60 msec | 1 | 0 |
  Maximum Post-Baseline Value : Increase from Baseline QTcF Interval > 60 msec: number analyzed (Participants) | 7 | 5 | 0
  Maximum Post-Baseline Value : Increase from Baseline QTcF Interval > 60 msec | 0 | 0 |
  Maximum Post-Baseline Value : Missing: number analyzed (Participants) | 7 | 5 | 0
  Maximum Post-Baseline Value : Missing | 0 | 1 |
  Last Post-Baseline Value : QTcF Interval > 450 - 480 msec: number analyzed (Participants) | 7 | 5 | 0
  Last Post-Baseline Value : QTcF Interval > 450 - 480 msec | 0 | 0 |
  Last Post-Baseline Value : QTcF Interval > 480 - 500 msec: number analyzed (Participants) | 7 | 5 | 0
  Last Post-Baseline Value : QTcF Interval > 480 - 500 msec | 0 | 0 |
  Last Post-Baseline Value : QTcF Interval > 500 msec: number analyzed (Participants) | 7 | 5 | 0
  Last Post-Baseline Value : QTcF Interval > 500 msec | 0 | 0 |
  Last Post-Baseline Value : Increase from Baseline QTcF Interval > 30 - 60 msec: number analyzed (Participants) | 7 | 5 | 0
  Last Post-Baseline Value : Increase from Baseline QTcF Interval > 30 - 60 msec | 1 | 0 |
  Last Post-Baseline Value : Increase from Baseline QTcF Interval > 60 msec: number analyzed (Participants) | 7 | 5 | 0
  Last Post-Baseline Value : Increase from Baseline QTcF Interval > 60 msec | 0 | 0 |
  Last Post-Baseline Value : Missing: number analyzed (Participants) | 7 | 5 | 0
  Last Post-Baseline Value : Missing | 0 | 1 |

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Values Over Time in Liver Function Tests: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: as for outcome 4
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 13, 17, 21, 26, 52, End of Treatment (up to Week 25), Week 104/End of Trial
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  ALT Baseline : >= 3 x upper limit of normal (ULN) | 0 | 0 | 0
  ALT Baseline : >= 5 x ULN | 0 | 0 | 0
  ALT Baseline : >= 10 x ULN | 0 | 0 | 0
  ALT Baseline : >= 20 x ULN | 0 | 0 | 0
  ALT Baseline : Missing | 0 | 0 | 0
  ALT Week 1 : >= 3 x ULN | 2 | 2 | 0
  ALT Week 1 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 1 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 1 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 1 : Missing | 0 | 0 | 0
  ALT Week 2 : >= 3 x ULN: number analyzed (Participants) | 14 | 14 | 1
  ALT Week 2 : >= 3 x ULN | 1 | 0 | 0
  ALT Week 2 : >= 5 x ULN: number analyzed (Participants) | 14 | 14 | 1
  ALT Week 2 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 2 : >= 10 x ULN: number analyzed (Participants) | 14 | 14 | 1
  ALT Week 2 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 2 : >= 20 x ULN: number analyzed (Participants) | 14 | 14 | 1
  ALT Week 2 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  ALT Week 2 : Missing | 0 | 0 | 0
  ALT Week 3 : >= 3 x ULN: number analyzed (Participants) | 13 | 13 | 1
  ALT Week 3 : >= 3 x ULN | 0 | 1 | 0
  ALT Week 3 : >= 5 x ULN: number analyzed (Participants) | 13 | 13 | 1
  ALT Week 3 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 3 : >= 10 x ULN: number analyzed (Participants) | 13 | 13 | 1
  ALT Week 3 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 3 : >= 20 x ULN: number analyzed (Participants) | 13 | 13 | 1
  ALT Week 3 : >= 20 x ULN | 1 | 0 | 0
  ALT Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  ALT Week 3 : Missing | 0 | 0 | 0
  ALT Week 4 : >= 3 x ULN: number analyzed (Participants) | 12 | 12 | 1
  ALT Week 4 : >= 3 x ULN | 0 | 0 | 0
  ALT Week 4 : >= 5 x ULN: number analyzed (Participants) | 12 | 12 | 1
  ALT Week 4 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 4 : >= 10 x ULN: number analyzed (Participants) | 12 | 12 | 1
  ALT Week 4 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 4 : >= 20 x ULN: number analyzed (Participants) | 12 | 12 | 1
  ALT Week 4 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  ALT Week 4 : Missing | 0 | 0 | 0
  ALT Week 6 : >= 3 x ULN: number analyzed (Participants) | 11 | 9 | 1
  ALT Week 6 : >= 3 x ULN | 0 | 0 | 0
  ALT Week 6 : >= 5 x ULN: number analyzed (Participants) | 11 | 9 | 1
  ALT Week 6 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 6 : >= 10 x ULN: number analyzed (Participants) | 11 | 9 | 1
  ALT Week 6 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 6 : >= 20 x ULN: number analyzed (Participants) | 11 | 9 | 1
  ALT Week 6 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  ALT Week 6 : Missing | 0 | 0 | 0
  ALT Week 8 : >= 3 x ULN: number analyzed (Participants) | 10 | 8 | 1
  ALT Week 8 : >= 3 x ULN | 0 | 0 | 0
  ALT Week 8 : >= 5 x ULN: number analyzed (Participants) | 10 | 8 | 1
  ALT Week 8 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 8 : >= 10 x ULN: number analyzed (Participants) | 10 | 8 | 1
  ALT Week 8 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 8 : >= 20 x ULN: number analyzed (Participants) | 10 | 8 | 1
  ALT Week 8 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  ALT Week 8 : Missing | 0 | 0 | 0
  ALT Week 13 : >= 3 x ULN: number analyzed (Participants) | 8 | 8 | 1
  ALT Week 13 : >= 3 x ULN | 1 | 0 | 1
  ALT Week 13 : >= 5 x ULN: number analyzed (Participants) | 8 | 8 | 1
  ALT Week 13 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 13 : >= 10 x ULN: number analyzed (Participants) | 8 | 8 | 1
  ALT Week 13 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 13 : >= 20 x ULN: number analyzed (Participants) | 8 | 8 | 1
  ALT Week 13 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  ALT Week 13 : Missing | 1 | 0 | 0
  ALT Week 17 : >= 3 x ULN: number analyzed (Participants) | 7 | 7 | 1
  ALT Week 17 : >= 3 x ULN | 0 | 0 | 0
  ALT Week 17 : >= 5 x ULN: number analyzed (Participants) | 7 | 7 | 1
  ALT Week 17 : >= 5 x ULN | 0 | 0 | 0
  ALT Week 17 : >= 10 x ULN: number analyzed (Participants) | 7 | 7 | 1
  ALT Week 17 : >= 10 x ULN | 0 | 0 | 0
  ALT Week 17 : >= 20 x ULN: number analyzed (Participants) | 7 | 7 | 1
  ALT Week 17 : >= 20 x ULN | 0 | 0 | 0
  ALT Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  ALT Week 17 : Missing | 0 | 0 | 0
  ALT Week 21 : >= 3 x ULN: number analyzed (Participants) | 4 | 7 | 0
  ALT Week 21 : >= 3 x ULN | 0 | 0 |
  ALT Week 21 : >= 5 x ULN: number analyzed (Participants) | 4 | 7 | 0
  ALT Week 21 : >= 5 x ULN | 0 | 0 |
  ALT Week 21 : >= 10 x ULN: number analyzed (Participants) | 4 | 7 | 0
  ALT Week 21 : >= 10 x ULN | 0 | 0 |
  ALT Week 21 : >= 20 x ULN: number analyzed (Participants) | 4 | 7 | 0
  ALT Week 21 : >= 20 x ULN | 0 | 0 |
  ALT Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  ALT Week 21 : Missing | 0 | 0 |
  ALT Week 26 : >= 3 x ULN: number analyzed (Participants) | 4 | 5 | 0
  ALT Week 26 : >= 3 x ULN | 1 | 0 |
  ALT Week 26 : >= 5 x ULN: number analyzed (Participants) | 4 | 5 | 0
  ALT Week 26 : >= 5 x ULN | 0 | 0 |
  ALT Week 26 : >= 10 x ULN: number analyzed (Participants) | 4 | 5 | 0
  ALT Week 26 : >= 10 x ULN | 0 | 0 |
  ALT Week 26 : >= 20 x ULN: number analyzed (Participants) | 4 | 5 | 0
  ALT Week 26 : >= 20 x ULN | 0 | 0 |
  ALT Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  ALT Week 26 : Missing | 0 | 0 |
  ALT Week 52 : >= 3 x ULN: number analyzed (Participants) | 2 | 0 | 0
  ALT Week 52 : >= 3 x ULN | 0 |  |
  ALT Week 52 : >= 5 x ULN: number analyzed (Participants) | 2 | 0 | 0
  ALT Week 52 : >= 5 x ULN | 0 |  |
  ALT Week 52 : >= 10 x ULN: number analyzed (Participants) | 2 | 0 | 0
  ALT Week 52 : >= 10 x ULN | 0 |  |
  ALT Week 52 : >= 20 x ULN: number analyzed (Participants) | 2 | 0 | 0
  ALT Week 52 : >= 20 x ULN | 0 |  |
  ALT Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  ALT Week 52 : Missing | 0 |  |
  ALT End of Treatment : >= 3 x ULN: number analyzed (Participants) | 0 | 2 | 0
  ALT End of Treatment : >= 3 x ULN |  | 0 |
  ALT End of Treatment : >= 5 x ULN: number analyzed (Participants) | 0 | 2 | 0
  ALT End of Treatment : >= 5 x ULN |  | 0 |
  ALT End of Treatment : >= 10 x ULN: number analyzed (Participants) | 0 | 2 | 0
  ALT End of Treatment : >= 10 x ULN |  | 0 |
  ALT End of Treatment : >= 20 x ULN: number analyzed (Participants) | 0 | 2 | 0
  ALT End of Treatment : >= 20 x ULN |  | 0 |
  ALT End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  ALT End of Treatment : Missing |  | 0 |
  ALT Week 104/End of Trial : >= 3 x ULN: number analyzed (Participants) | 5 | 2 | 0
  ALT Week 104/End of Trial : >= 3 x ULN | 0 | 0 |
  ALT Week 104/End of Trial : >= 5 x ULN: number analyzed (Participants) | 5 | 2 | 0
  ALT Week 104/End of Trial : >= 5 x ULN | 0 | 1 |
  ALT Week 104/End of Trial : >= 10 x ULN: number analyzed (Participants) | 5 | 2 | 0
  ALT Week 104/End of Trial : >= 10 x ULN | 0 | 0 |
  ALT Week 104/End of Trial : >= 20 x ULN: number analyzed (Participants) | 5 | 2 | 0
  ALT Week 104/End of Trial : >= 20 x ULN | 0 | 0 |
  ALT Week 104/End of Trial : Missing: number analyzed (Participants) | 5 | 2 | 0
  ALT Week 104/End of Trial : Missing | 0 | 0 |
  ALT Minimum Post-Baseline Value : >= 3 x ULN | 0 | 1 | 0
  ALT Minimum Post-Baseline Value : >= 5 x ULN | 0 | 0 | 0
  ALT Minimum Post-Baseline Value : >= 10 x ULN | 0 | 0 | 0
  ALT Minimum Post-Baseline Value : >= 20 x ULN | 0 | 0 | 0
  ALT Minimum Post-Baseline Value : Missing | 0 | 0 | 0
  ALT Maximum Post-Baseline Value : >= 3 x ULN | 3 | 3 | 0
  ALT Maximum Post-Baseline Value : >= 5 x ULN | 1 | 1 | 1
  ALT Maximum Post-Baseline Value : >= 10 x ULN | 0 | 0 | 0
  ALT Maximum Post-Baseline Value : >= 20 x ULN | 1 | 0 | 0
  ALT Maximum Post-Baseline Value : Missing | 0 | 0 | 0
  ALT Last Post-Baseline Value : >= 3 x ULN | 1 | 0 | 0
  ALT Last Post-Baseline Value : >= 5 x ULN | 0 | 1 | 1
  ALT Last Post-Baseline Value : >= 10 x ULN | 0 | 0 | 0
  ALT Last Post-Baseline Value : >= 20 x ULN | 1 | 0 | 0
  ALT Last Post-Baseline Value : Missing | 0 | 0 | 0
  AST Baseline : >= 3 x ULN | 0 | 0 | 0
  AST Baseline : >= 5 x ULN | 0 | 0 | 0
  AST Baseline : >= 10 x ULN | 0 | 0 | 0
  AST Baseline : >= 20 x ULN | 0 | 0 | 0
  AST Baseline : Missing | 0 | 0 | 0
  AST Week 1 : >= 3 x ULN | 0 | 0 | 0
  AST Week 1 : >= 5 x ULN | 0 | 1 | 0
  AST Week 1 : >= 10 x ULN | 0 | 0 | 0
  AST Week 1 : >= 20 x ULN | 0 | 0 | 0
  AST Week 1 : Missing | 0 | 0 | 0
  AST Week 2 : >= 3 x ULN: number analyzed (Participants) | 14 | 14 | 1
  AST Week 2 : >= 3 x ULN | 0 | 0 | 0
  AST Week 2 : >= 5 x ULN: number analyzed (Participants) | 14 | 14 | 1
  AST Week 2 : >= 5 x ULN | 0 | 0 | 0
  AST Week 2 : >= 10 x ULN: number analyzed (Participants) | 14 | 14 | 1
  AST Week 2 : >= 10 x ULN | 0 | 0 | 0
  AST Week 2 : >= 20 x ULN: number analyzed (Participants) | 14 | 14 | 1
  AST Week 2 : >= 20 x ULN | 0 | 0 | 0
  AST Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  AST Week 2 : Missing | 1 | 0 | 0
  AST Week 3 : >= 3 x ULN: number analyzed (Participants) | 13 | 13 | 1
  AST Week 3 : >= 3 x ULN | 0 | 0 | 0
  AST Week 3 : >= 5 x ULN: number analyzed (Participants) | 13 | 13 | 1
  AST Week 3 : >= 5 x ULN | 0 | 0 | 0
  AST Week 3 : >= 10 x ULN: number analyzed (Participants) | 13 | 13 | 1
  AST Week 3 : >= 10 x ULN | 0 | 0 | 0
  AST Week 3 : >= 20 x ULN: number analyzed (Participants) | 13 | 13 | 1
  AST Week 3 : >= 20 x ULN | 1 | 0 | 0
  AST Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  AST Week 3 : Missing | 0 | 0 | 0
  AST Week 4 : >= 3 x ULN: number analyzed (Participants) | 12 | 12 | 1
  AST Week 4 : >= 3 x ULN | 0 | 0 | 0
  AST Week 4 : >= 5 x ULN: number analyzed (Participants) | 12 | 12 | 1
  AST Week 4 : >= 5 x ULN | 0 | 0 | 0
  AST Week 4 : >= 10 x ULN: number analyzed (Participants) | 12 | 12 | 1
  AST Week 4 : >= 10 x ULN | 0 | 0 | 0
  AST Week 4 : >= 20 x ULN: number analyzed (Participants) | 12 | 12 | 1
  AST Week 4 : >= 20 x ULN | 0 | 0 | 0
  AST Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  AST Week 4 : Missing | 0 | 0 | 0
  AST Week 6 : >= 3 x ULN: number analyzed (Participants) | 11 | 9 | 1
  AST Week 6 : >= 3 x ULN | 0 | 0 | 0
  AST Week 6 : >= 5 x ULN: number analyzed (Participants) | 11 | 9 | 1
  AST Week 6 : >= 5 x ULN | 0 | 0 | 0
  AST Week 6 : >= 10 x ULN: number analyzed (Participants) | 11 | 9 | 1
  AST Week 6 : >= 10 x ULN | 0 | 0 | 0
  AST Week 6 : >= 20 x ULN: number analyzed (Participants) | 11 | 9 | 1
  AST Week 6 : >= 20 x ULN | 0 | 0 | 0
  AST Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  AST Week 6 : Missing | 0 | 0 | 0
  AST Week 8 : >= 3 x ULN: number analyzed (Participants) | 10 | 8 | 1
  AST Week 8 : >= 3 x ULN | 0 | 0 | 0
  AST Week 8 : >= 5 x ULN: number analyzed (Participants) | 10 | 8 | 1
  AST Week 8 : >= 5 x ULN | 0 | 0 | 0
  AST Week 8 : >= 10 x ULN: number analyzed (Participants) | 10 | 8 | 1
  AST Week 8 : >= 10 x ULN | 0 | 0 | 0
  AST Week 8 : >= 20 x ULN: number analyzed (Participants) | 10 | 8 | 1
  AST Week 8 : >= 20 x ULN | 0 | 0 | 0
  AST Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  AST Week 8 : Missing | 0 | 0 | 0
  AST Week 13 : >= 3 x ULN: number analyzed (Participants) | 8 | 8 | 1
  AST Week 13 : >= 3 x ULN | 1 | 0 | 0
  AST Week 13 : >= 5 x ULN: number analyzed (Participants) | 8 | 8 | 1
  AST Week 13 : >= 5 x ULN | 0 | 0 | 0
  AST Week 13 : >= 10 x ULN: number analyzed (Participants) | 8 | 8 | 1
  AST Week 13 : >= 10 x ULN | 0 | 0 | 0
  AST Week 13 : >= 20 x ULN: number analyzed (Participants) | 8 | 8 | 1
  AST Week 13 : >= 20 x ULN | 0 | 0 | 0
  AST Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  AST Week 13 : Missing | 1 | 0 | 0
  AST Week 17 : >= 3 x ULN: number analyzed (Participants) | 7 | 7 | 1
  AST Week 17 : >= 3 x ULN | 0 | 0 | 0
  AST Week 17 : >= 5 x ULN: number analyzed (Participants) | 7 | 7 | 1
  AST Week 17 : >= 5 x ULN | 0 | 0 | 0
  AST Week 17 : >= 10 x ULN: number analyzed (Participants) | 7 | 7 | 1
  AST Week 17 : >= 10 x ULN | 0 | 0 | 0
  AST Week 17 : >= 20 x ULN: number analyzed (Participants) | 7 | 7 | 1
  AST Week 17 : >= 20 x ULN | 0 | 0 | 0
  AST Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  AST Week 17 : Missing | 0 | 0 | 0
  AST Week 21 : >= 3 x ULN: number analyzed (Participants) | 4 | 7 | 0
  AST Week 21 : >= 3 x ULN | 0 | 0 |
  AST Week 21 : >= 5 x ULN: number analyzed (Participants) | 4 | 7 | 0
  AST Week 21 : >= 5 x ULN | 0 | 0 |
  AST Week 21 : >= 10 x ULN: number analyzed (Participants) | 4 | 7 | 0
  AST Week 21 : >= 10 x ULN | 0 | 0 |
  AST Week 21 : >= 20 x ULN: number analyzed (Participants) | 4 | 7 | 0
  AST Week 21 : >= 20 x ULN | 0 | 0 |
  AST Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  AST Week 21 : Missing | 0 | 0 |
  AST Week 26 : >= 3 x ULN: number analyzed (Participants) | 4 | 5 | 0
  AST Week 26 : >= 3 x ULN | 1 | 0 |
  AST Week 26 : >= 5 x ULN: number analyzed (Participants) | 4 | 5 | 0
  AST Week 26 : >= 5 x ULN | 0 | 0 |
  AST Week 26 : >= 10 x ULN: number analyzed (Participants) | 4 | 5 | 0
  AST Week 26 : >= 10 x ULN | 0 | 0 |
  AST Week 26 : >= 20 x ULN: number analyzed (Participants) | 4 | 5 | 0
  AST Week 26 : >= 20 x ULN | 0 | 0 |
  AST Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  AST Week 26 : Missing | 0 | 0 |
  AST Week 52 : >= 3 x ULN: number analyzed (Participants) | 2 | 0 | 0
  AST Week 52 : >= 3 x ULN | 0 |  |
  AST Week 52 : >= 5 x ULN: number analyzed (Participants) | 2 | 0 | 0
  AST Week 52 : >= 5 x ULN | 0 |  |
  AST Week 52 : >= 10 x ULN: number analyzed (Participants) | 2 | 0 | 0
  AST Week 52 : >= 10 x ULN | 0 |  |
  AST Week 52 : >= 20 x ULN: number analyzed (Participants) | 2 | 0 | 0
  AST Week 52 : >= 20 x ULN | 0 |  |
  AST Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  AST Week 52 : Missing | 0 |  |
  AST End of Treatment : >= 3 x ULN: number analyzed (Participants) | 0 | 2 | 0
  AST End of Treatment : >= 3 x ULN |  | 0 |
  AST End of Treatment : >= 5 x ULN: number analyzed (Participants) | 0 | 2 | 0
  AST End of Treatment : >= 5 x ULN |  | 0 |
  AST End of Treatment : >= 10 x ULN: number analyzed (Participants) | 0 | 2 | 0
  AST End of Treatment : >= 10 x ULN |  | 0 |
  AST End of Treatment : >= 20 x ULN: number analyzed (Participants) | 0 | 2 | 0
  AST End of Treatment : >= 20 x ULN |  | 0 |
  AST End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  AST End of Treatment : Missing |  | 0 |
  AST Week 104/End of Trial : >= 3 x ULN: number analyzed (Participants) | 5 | 2 | 0
  AST Week 104/End of Trial : >= 3 x ULN | 0 | 0 |
  AST Week 104/End of Trial : >= 5 x ULN: number analyzed (Participants) | 5 | 2 | 0
  AST Week 104/End of Trial : >= 5 x ULN | 0 | 0 |
  AST Week 104/End of Trial : >= 10 x ULN: number analyzed (Participants) | 5 | 2 | 0
  AST Week 104/End of Trial : >= 10 x ULN | 0 | 1 |
  AST Week 104/End of Trial : >= 20 x ULN: number analyzed (Participants) | 5 | 2 | 0
  AST Week 104/End of Trial : >= 20 x ULN | 0 | 0 |
  AST Week 104/End of Trial : Missing: number analyzed (Participants) | 5 | 2 | 0
  AST Week 104/End of Trial : Missing | 0 | 0 |
  AST Minimum Post-Baseline Value : >= 3 x ULN | 0 | 0 | 0
  AST Minimum Post-Baseline Value : >= 5 x ULN | 0 | 1 | 0
  AST Minimum Post-Baseline Value : >= 10 x ULN | 0 | 0 | 0
  AST Minimum Post-Baseline Value : >= 20 x ULN | 0 | 0 | 0
  AST Minimum Post-Baseline Value : Missing | 0 | 0 | 0
  AST Maximum Post-Baseline Value : >= 3 x ULN | 2 | 1 | 1
  AST Maximum Post-Baseline Value : >= 5 x ULN | 0 | 0 | 0
  AST Maximum Post-Baseline Value : >= 10 x ULN | 0 | 1 | 0
  AST Maximum Post-Baseline Value : >= 20 x ULN | 1 | 0 | 0
  AST Maximum Post-Baseline Value : Missing | 0 | 0 | 0
  AST Last Post-Baseline Value : >= 3 x ULN | 1 | 0 | 1
  AST Last Post-Baseline Value : >= 5 x ULN | 0 | 0 | 0
  AST Last Post-Baseline Value : >= 10 x ULN | 0 | 1 | 0
  AST Last Post-Baseline Value : >= 20 x ULN | 1 | 0 | 0
  AST Last Post-Baseline Value : Missing | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Values Over Time in Liver Function Tests: Total Bilirubin
Description: as for outcome 4
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 52, End of Treatment (up to Week 25), Week 104/End of Trial
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Baseline : >= 2 x Upper Limit of Normal (ULN) | 0 | 0 | 0
  Baseline : Missing | 0 | 0 | 0
  Week 1 : >= 2 x ULN | 1 | 0 | 0
  Week 1 : Missing | 0 | 0 | 0
  Week 2 : >= 2 x ULN: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : >= 2 x ULN | 1 | 1 | 0
  Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Missing | 0 | 0 | 0
  Week 3 : >= 2 x ULN: number analyzed (Participants) | 13 | 13 | 1
  Week 3 : >= 2 x ULN | 1 | 0 | 0
  Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  Week 3 : Missing | 0 | 0 | 0
  Week 4 : >= 2 x ULN: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : >= 2 x ULN | 0 | 0 | 0
  Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Missing | 0 | 0 | 0
  Week 5 : >= 2 x ULN: number analyzed (Participants) | 12 | 10 | 1
  Week 5 : >= 2 x ULN | 0 | 0 | 0
  Week 5 : Missing: number analyzed (Participants) | 12 | 10 | 1
  Week 5 : Missing | 0 | 0 | 0
  Week 6 : >= 2 x ULN: number analyzed (Participants) | 11 | 9 | 1
  Week 6 : >= 2 x ULN | 0 | 0 | 0
  Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  Week 6 : Missing | 0 | 0 | 0
  Week 7 : >= 2 x ULN: number analyzed (Participants) | 9 | 9 | 1
  Week 7 : >= 2 x ULN | 0 | 0 | 0
  Week 7 : Missing: number analyzed (Participants) | 9 | 9 | 1
  Week 7 : Missing | 0 | 0 | 0
  Week 8 : >= 2 x ULN: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : >= 2 x ULN | 0 | 0 | 0
  Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Missing | 0 | 0 | 0
  Week 9 : >= 2 x ULN: number analyzed (Participants) | 4 | 6 | 0
  Week 9 : >= 2 x ULN | 0 | 0 |
  Week 9 : Missing: number analyzed (Participants) | 4 | 6 | 0
  Week 9 : Missing | 0 | 0 |
  Week 10 : >= 2 x ULN: number analyzed (Participants) | 4 | 6 | 0
  Week 10 : >= 2 x ULN | 0 | 0 |
  Week 10 : Missing: number analyzed (Participants) | 4 | 6 | 0
  Week 10 : Missing | 0 | 0 |
  Week 11 : >= 2 x ULN: number analyzed (Participants) | 4 | 6 | 0
  Week 11 : >= 2 x ULN | 0 | 0 |
  Week 11 : Missing: number analyzed (Participants) | 4 | 6 | 0
  Week 11 : Missing | 0 | 0 |
  Week 12 : >= 2 x ULN: number analyzed (Participants) | 2 | 5 | 0
  Week 12 : >= 2 x ULN | 0 | 0 |
  Week 12 : Missing: number analyzed (Participants) | 2 | 5 | 0
  Week 12 : Missing | 0 | 0 |
  Week 13 : >= 2 x ULN: number analyzed (Participants) | 8 | 8 | 1
  Week 13 : >= 2 x ULN | 0 | 0 | 0
  Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  Week 13 : Missing | 1 | 0 | 0
  Week 14 : >= 2 x ULN: number analyzed (Participants) | 0 | 3 | 0
  Week 14 : >= 2 x ULN |  | 0 |
  Week 14 : Missing: number analyzed (Participants) | 0 | 3 | 0
  Week 14 : Missing |  | 0 |
  Week 15 : >= 2 x ULN: number analyzed (Participants) | 0 | 3 | 0
  Week 15 : >= 2 x ULN |  | 0 | 0
  Week 15 : Missing: number analyzed (Participants) | 0 | 3 | 0
  Week 15 : Missing |  | 0 | 0
  Week 16 : >= 2 x ULN: number analyzed (Participants) | 0 | 3 | 0
  Week 16 : >= 2 x ULN |  | 0 |
  Week 16 : Missing: number analyzed (Participants) | 0 | 3 | 0
  Week 16 : Missing |  | 0 |
  Week 17 : >= 2 x ULN: number analyzed (Participants) | 7 | 7 | 1
  Week 17 : >= 2 x ULN | 0 | 0 | 0
  Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  Week 17 : Missing | 0 | 0 | 0
  Week 18 : >= 2 x ULN: number analyzed (Participants) | 0 | 2 | 1
  Week 18 : >= 2 x ULN |  | 0 | 0
  Week 18 : Missing: number analyzed (Participants) | 0 | 2 | 1
  Week 18 : Missing |  | 0 | 0
  Week 19 : >= 2 x ULN: number analyzed (Participants) | 0 | 2 | 1
  Week 19 : >= 2 x ULN |  | 0 | 1
  Week 19 : Missing: number analyzed (Participants) | 0 | 2 | 1
  Week 19 : Missing |  | 0 | 0
  Week 20 : >= 2 x ULN: number analyzed (Participants) | 0 | 2 | 0
  Week 20 : >= 2 x ULN |  | 0 |
  Week 20 : Missing: number analyzed (Participants) | 0 | 2 | 0
  Week 20 : Missing |  | 0 |
  Week 21 : >= 2 x ULN: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : >= 2 x ULN | 0 | 0 |
  Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Missing | 0 | 0 |
  Week 22 : >= 2 x ULN: number analyzed (Participants) | 0 | 2 | 0
  Week 22 : >= 2 x ULN |  | 0 |
  Week 22 : Missing: number analyzed (Participants) | 0 | 2 | 0
  Week 22 : Missing |  | 0 |
  Week 23 : >= 2 x ULN: number analyzed (Participants) | 0 | 1 | 0
  Week 23 : >= 2 x ULN |  | 0 |
  Week 23 : Missing: number analyzed (Participants) | 0 | 1 | 0
  Week 23 : Missing |  | 0 |
  Week 24 : >= 2 x ULN: number analyzed (Participants) | 0 | 1 | 0
  Week 24 : >= 2 x ULN |  | 0 |
  Week 24 : Missing: number analyzed (Participants) | 0 | 1 | 0
  Week 24 : Missing |  | 0 |
  Week 25 : >= 2 x ULN: number analyzed (Participants) | 0 | 1 | 0
  Week 25 : >= 2 x ULN |  | 0 |
  Week 25 : Missing: number analyzed (Participants) | 0 | 1 | 0
  Week 25 : Missing |  | 0 |
  Week 26 : >= 2 x ULN: number analyzed (Participants) | 4 | 5 | 0
  Week 26 : >= 2 x ULN | 0 | 0 |
  Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  Week 26 : Missing | 0 | 0 |
  Week 52 : >= 2 x ULN: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : >= 2 x ULN | 0 |  |
  Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : Missing | 0 |  |
  End of Treatment : >= 2 x ULN: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : >= 2 x ULN |  | 0 |
  End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Missing |  | 0 |
  Week 104/End of Trial : >= 2 x ULN: number analyzed (Participants) | 5 | 2 | 0
  Week 104/End of Trial : >= 2 x ULN | 0 | 0 |
  Week 104/End of Trial : Missing: number analyzed (Participants) | 5 | 2 | 0
  Week 104/End of Trial : Missing | 0 | 0 |
  Minimum Post-Baseline Value : >= 2 x ULN | 1 | 0 | 0
  Minimum Post-Baseline Value : Missing | 0 | 0 | 0
  Maximum Post-Baseline Value : >= 2 x ULN | 1 | 1 | 1
  Maximum Post-Baseline Value : Missing | 0 | 0 | 0
  Last Post-Baseline Value : >= 2 x ULN | 1 | 0 | 1
  Last Post-Baseline Value : Missing | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Values Over Time in Liver Function Tests: Potential Hy's Law Cases
Description: Potential Hy's Law cases were defined as ALT or AST >= 3 x ULN AND total bilirubin >= 2 x ULN AND alkaline phosphatase (ALP) <= 2 x ULN at the same visit.
  Baseline is defined as the last measurement prior to the first dose of apraglutide.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 13, 17, 21, 26, 52, End of Treatment (up to Week 25), Week 104/End of Trial
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Baseline : Potential Hy's Law Cases | 0 | 0 | 0
  Baseline : Missing | 0 | 0 | 0
  Week 1 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 1 : Missing | 0 | 2 | 0
  Week 2 : Potential Hy's Law Cases: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 2 : Missing: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Missing | 1 | 0 | 0
  Week 3 : Potential Hy's Law Cases: number analyzed (Participants) | 13 | 13 | 1
  Week 3 : Potential Hy's Law Cases | 1 | 0 | 0
  Week 3 : Missing: number analyzed (Participants) | 13 | 13 | 1
  Week 3 : Missing | 0 | 0 | 0
  Week 4 : Potential Hy's Law Cases: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 4 : Missing: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Missing | 0 | 0 | 0
  Week 6 : Potential Hy's Law Cases: number analyzed (Participants) | 11 | 9 | 1
  Week 6 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 6 : Missing: number analyzed (Participants) | 11 | 9 | 1
  Week 6 : Missing | 1 | 0 | 0
  Week 8 : Potential Hy's Law Cases: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 8 : Missing: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Missing | 1 | 0 | 0
  Week 13 : Potential Hy's Law Cases: number analyzed (Participants) | 8 | 8 | 1
  Week 13 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 13 : Missing: number analyzed (Participants) | 8 | 8 | 1
  Week 13 : Missing | 1 | 0 | 0
  Week 17 : Potential Hy's Law Cases: number analyzed (Participants) | 7 | 7 | 1
  Week 17 : Potential Hy's Law Cases | 0 | 0 | 0
  Week 17 : Missing: number analyzed (Participants) | 7 | 7 | 1
  Week 17 : Missing | 0 | 0 | 0
  Week 21 : Potential Hy's Law Cases: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Potential Hy's Law Cases | 0 | 0 |
  Week 21 : Missing: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Missing | 0 | 0 |
  Week 26 : Potential Hy's Law Cases: number analyzed (Participants) | 4 | 5 | 0
  Week 26 : Potential Hy's Law Cases | 0 | 0 |
  Week 26 : Missing: number analyzed (Participants) | 4 | 5 | 0
  Week 26 : Missing | 0 | 0 |
  Week 52 : Potential Hy's Law Cases: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : Potential Hy's Law Cases | 0 |  |
  Week 52 : Missing: number analyzed (Participants) | 2 | 0 | 0
  Week 52 : Missing | 0 |  |
  End of Treatment : Potential Hy's Law Cases: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Potential Hy's Law Cases |  | 0 |
  End of Treatment : Missing: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Missing |  | 0 |
  Week 104/End of Trial : Potential Hy's Law Cases: number analyzed (Participants) | 5 | 2 | 0
  Week 104/End of Trial : Potential Hy's Law Cases | 0 | 0 |
  Week 104/End of Trial : Missing: number analyzed (Participants) | 5 | 2 | 0
  Week 104/End of Trial : Missing | 0 | 0 |

8. Primary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) Over Time
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 13, 17, 21, 26, 52, End of Treatment (up to Week 25), Week 104/End of Trial
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Baseline : Screening = Negative | 14 | 15 | 1
  Baseline : Screening = Potentially Positive | 1 | 0 | 0
  Baseline : Confirmation = Negative Immunodepletion | 1 | 0 | 0
  Baseline : Confirmation = Positive | 0 | 0 | 0
  Week 1 : Screening = Negative | 14 | 14 | 1
  Week 1 : Screening = Potentially Positive | 1 | 1 | 0
  Week 1 : Confirmation = Negative Immunodepletion | 1 | 1 | 0
  Week 1 : Confirmation = Positive | 0 | 0 | 0
  Week 2 : Screening = Negative: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Screening = Negative | 14 | 14 | 1
  Week 2 : Screening = Potentially Positive: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Screening = Potentially Positive | 0 | 0 | 0
  Week 2 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Confirmation = Negative Immunodepletion | 0 | 0 | 0
  Week 2 : Confirmation = Positive: number analyzed (Participants) | 14 | 14 | 1
  Week 2 : Confirmation = Positive | 0 | 0 | 0
  Week 4 : Screening = Negative: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Screening = Negative | 12 | 11 | 1
  Week 4 : Screening = Potentially Positive: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Screening = Potentially Positive | 0 | 1 | 0
  Week 4 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Confirmation = Negative Immunodepletion | 0 | 1 | 0
  Week 4 : Confirmation = Positive: number analyzed (Participants) | 12 | 12 | 1
  Week 4 : Confirmation = Positive | 0 | 0 | 0
  Week 8 : Screening = Negative: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Screening = Negative | 10 | 8 | 1
  Week 8 : Screening = Potentially Positive: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Screening = Potentially Positive | 0 | 0 | 0
  Week 8 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Confirmation = Negative Immunodepletion | 0 | 0 | 0
  Week 8 : Confirmation = Positive: number analyzed (Participants) | 10 | 8 | 1
  Week 8 : Confirmation = Positive | 0 | 0 | 0
  Week 13 : Screening = Negative: number analyzed (Participants) | 7 | 8 | 1
  Week 13 : Screening = Negative | 7 | 8 | 1
  Week 13 : Screening = Potentially Positive: number analyzed (Participants) | 7 | 8 | 1
  Week 13 : Screening = Potentially Positive | 0 | 0 | 0
  Week 13 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 7 | 8 | 1
  Week 13 : Confirmation = Negative Immunodepletion | 0 | 0 | 0
  Week 13 : Confirmation = Positive: number analyzed (Participants) | 7 | 8 | 1
  Week 13 : Confirmation = Positive | 0 | 0 | 0
  Week 17 : Screening = Negative: number analyzed (Participants) | 7 | 6 | 1
  Week 17 : Screening = Negative | 6 | 6 | 1
  Week 17 : Screening = Potentially Positive: number analyzed (Participants) | 7 | 6 | 1
  Week 17 : Screening = Potentially Positive | 1 | 0 | 0
  Week 17 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 7 | 6 | 1
  Week 17 : Confirmation = Negative Immunodepletion | 1 | 0 | 0
  Week 17 : Confirmation = Positive: number analyzed (Participants) | 7 | 6 | 1
  Week 17 : Confirmation = Positive | 0 | 0 | 0
  Week 21 : Screening = Negative: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Screening = Negative | 4 | 7 |
  Week 21 : Screening = Potentially Positive: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Screening = Potentially Positive | 0 | 0 |
  Week 21 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Confirmation = Negative Immunodepletion | 0 | 0 |
  Week 21 : Confirmation = Positive: number analyzed (Participants) | 4 | 7 | 0
  Week 21 : Confirmation = Positive | 0 | 0 |
  Week 52 : Screening = Negative: number analyzed (Participants) | 2 | 2 | 0
  Week 52 : Screening = Negative | 2 | 2 |
  Week 52 : Screening = Potentially Positive: number analyzed (Participants) | 2 | 2 | 0
  Week 52 : Screening = Potentially Positive | 0 | 0 |
  Week 52 : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 2 | 2 | 0
  Week 52 : Confirmation = Negative Immunodepletion | 0 | 2 |
  Week 52 : Confirmation = Positive: number analyzed (Participants) | 2 | 2 | 0
  Week 52 : Confirmation = Positive | 0 | 0 |
  End of Treatment : Screening = Negative: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Screening = Negative |  | 2 |
  End of Treatment : Screening = Potentially Positive: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Screening = Potentially Positive |  | 0 |
  End of Treatment : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Confirmation = Negative Immunodepletion |  | 0 |
  End of Treatment : Confirmation = Positive: number analyzed (Participants) | 0 | 2 | 0
  End of Treatment : Confirmation = Positive |  | 0 |
  Week 104/End of Trial : Screening = Negative: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Screening = Negative | 3 | 1 |
  Week 104/End of Trial : Screening = Potentially Positive: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Screening = Potentially Positive | 0 | 0 |
  Week 104/End of Trial : Confirmation = Negative Immunodepletion: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Confirmation = Negative Immunodepletion | 0 | 0 |
  Week 104/End of Trial : Confirmation = Positive: number analyzed (Participants) | 3 | 1 | 0
  Week 104/End of Trial : Confirmation = Positive | 0 | 0 |
  Last Post-Baseline Value : Screening = Negative | 14 | 14 | 1
  Last Post-Baseline Value : Screening = Potentially Positive | 1 | 1 | 0
  Last Post-Baseline Value : Confirmation = Negative Immunodepletion | 1 | 3 | 0
  Last Post-Baseline Value : Confirmation = Positive | 0 | 0 | 0

9. Primary Outcome: Shift Table From Baseline to Worst Post-Treatment (WPT) Physical Examinations
Time Frame: Baseline (BL), up to Week 104/End of Treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 8 | 9 | 1
Participants
  BL Abnormal, clinically significant (CS) : WPT Abnormal, CS | 4 | 3 | 0
  BL Abnormal, CS : WPT Abnormal, Not Clinically Significant (NCS): number analyzed (Participants) | 6 | 6 | 0
  BL Abnormal, CS : WPT Abnormal, Not Clinically Significant (NCS) | 0 | 0 |
  BL Abnormal, CS : WPT Normal: number analyzed (Participants) | 1 | 0 | 0
  BL Abnormal, CS : WPT Normal | 0 |  |
  BL Abnormal, CS : WPT Missing: number analyzed (Participants) | 0 | 0 | 0
  BL Abnormal, NCS : WPT Abnormal, CS | 3 | 5 | 1
  BL Abnormal, NCS : WPT Abnormal, NCS: number analyzed (Participants) | 6 | 6 | 0
  BL Abnormal, NCS : WPT Abnormal, NCS | 4 | 3 |
  BL Abnormal, NCS : WPT Normal: number analyzed (Participants) | 1 | 0 | 0
  BL Abnormal, NCS : WPT Normal | 1 |  |
  BL Abnormal, NCS : WPT Missing: number analyzed (Participants) | 0 | 0 | 0
  BL Normal : WPT Abnormal, CS | 1 | 1 | 0
  BL Normal : WPT Abnormal, NCS: number analyzed (Participants) | 6 | 6 | 0
  BL Normal : WPT Abnormal, NCS | 2 | 2 |
  BL Normal : WPT Normal: number analyzed (Participants) | 1 | 0 | 0
  BL Normal : WPT Normal | 0 |  |
  BL Normal : WPT Missing: number analyzed (Participants) | 0 | 0 | 0
  BL Missing : WPT Abnormal, CS: number analyzed (Participants) | 8 | 9 | 0
  BL Missing : WPT Abnormal, CS | 0 | 0 |
  BL Missing : WPT Abnormal, NCS: number analyzed (Participants) | 6 | 6 | 0
  BL Missing : WPT Abnormal, NCS | 0 | 1 |
  BL Missing : WPT Normal: number analyzed (Participants) | 1 | 0 | 0
  BL Missing : WPT Normal | 0 |  |
  BL Missing : WPT Missing: number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Overall Response Rate at Day 56 on the Lower Gastrointestinal (GI) Tract Mount Sinai aGVHD International Consortium (MAGIC) Stage
Description: Overall response rate at Day 56 on the lower GI tract MAGIC stage is defined as the percentage of participants with complete response (CR) or partial response (PR) on the lower GI tract MAGIC stage at Day 56. Lower GI (Stool Output/Day) MAGIC Stages are 0: <500 mL/day or <3/episodes/day; 1: 500-999 mL/day or 3-4/episodes/day; 2: 1000-1500 mL/day or 5-7/episodes/day; 3: >1500 mL/day or >7/episodes/day; 4: Severe abdominal pain with or without ileus or grossly bloody stool (regardless of volume).
  CR: Score of 0 in lower GI tract MAGIC stage that indicates complete resolution of all signs and symptoms of aGVHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGVHD. PR: Improvement of one stage in lower GI tract MAGIC stage without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response, or non-response of aGVHD.
Time Frame: Day 56
Population: Full Analysis Set: all enrolled participants
Measure: Number; unit: percentage of participants
Groups:
- Apraglutide High Dose: High-dose, weight-based apraglutide SC injections (5 to 10 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight of more than 50.0 kg.
- Apraglutide Standard Dose: Standard-dose apraglutide SC injections (2.5 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight between 40.0 kg to 49.9 kg.
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants | 53.3 | 46.7 | 100

11. Secondary Outcome: Overall Response Rate Over Time on the Lower GI Tract MAGIC Stage
Description: Overall response rate on the lower GI tract MAGIC stage is defined as the percentage of participants with CR or PR on the lower GI tract MAGIC stage at given time points. Lower GI (Stool Output/Day) MAGIC Stages are 0: <500 mL/day or <3/episodes/day; 1: 500-999 mL/day or 3-4/episodes/day; 2: 1000-1500 mL/day or 5-7/episodes/day; 3: >1500 mL/day or >7/episodes/day; 4: Severe abdominal pain with or without ileus or grossly bloody stool (regardless of volume).
  CR: Score of 0 in lower GI tract MAGIC stage that indicates complete resolution of all signs and symptoms of aGVHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGVHD. PR: Improvement of one stage in lower GI tract MAGIC stage without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response, or non-response of aGVHD.
Time Frame: Days 14, 28, 56, 91, 119, 147, and 182
Population: Full Analysis Set: all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants
  Day 14 | 53.3 [26.6 to 78.7] | 66.7 [38.4 to 88.2] | 100 [2.5 to 100]
  Day 28 | 66.7 [38.4 to 88.2] | 40.0 [16.3 to 67.7] | 100 [2.5 to 100]
  Day 56 | 53.3 [26.6 to 78.7] | 46.7 [21.3 to 73.4] | 100 [2.5 to 100]
  Day 91 | 46.7 [21.3 to 73.4] | 46.7 [21.3 to 73.4] | 100 [2.5 to 100]
  Day 119 | 40.0 [16.3 to 67.7] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]
  Day 147 | 26.7 [7.8 to 55.1] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]
  Day 182 | 26.7 [7.8 to 55.1] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]

12. Secondary Outcome: Overall Response Rate Over Time on the Total MAGIC Stage
Description: Overall response rate on Total MAGIC staging for each of the 4 evaluable organs of skin, lower and upper GI tract, and liver is defined as the percentage of participants with CR or PR on the total MAGIC stage. Staging values range from 0 to 4, with higher number indicating a worse state of disease. (For complete staging criteria, see: Harris AC, et al. Biol Blood Marrow Transplant. 2016;22(1):4-10.)
  CR: A score of 0 for the aGVHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGVHD in all 4 evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGVHD. PR: An improvement of one stage in one or more evaluable organs involved with aGVHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response, or non-response of aGVHD.
Time Frame: Days 14, 28, 56, 91, 119, 147, and 182
Population: Full Analysis Set: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants
  Day 14 | 53.3 [26.6 to 78.7] | 53.3 [26.6 to 78.7] | 100 [2.5 to 100]
  Day 28 | 66.7 [38.4 to 88.2] | 46.7 [21.3 to 73.4] | 100 [2.5 to 100]
  Day 56 | 53.3 [26.6 to 78.7] | 46.7 [21.3 to 73.4] | 100 [2.5 to 100]
  Day 91 | 40.0 [16.3 to 67.7] | 46.7 [21.3 to 73.4] | 100 [2.5 to 100]
  Day 119 | 33.3 [11.8 to 61.6] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]
  Day 147 | 26.7 [7.8 to 55.1] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]
  Day 182 | 26.7 [7.8 to 55.1] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]

13. Secondary Outcome: Durable Overall Response Rates on the Lower GI and Total MAGIC Score From Day 28 to Day 56
Description: Durable overall response rate on the Lower GI MAGIC Score from Day 28 to Day 56 is defined as the percentage of participants who had a response (either CR responder or PR responder, see Outcome Measure 10 description for details) on the lower GI at Day 28 and remain a CR responder or PR responder on the lower GI at Day 56.
  Durable overall response rate from Day 28 to Day 56 on the Total MAGIC Score is defined as the percentage of participants who had a response (either CR responder or PR responder, see Outcome Measure 12 description for details) on the total MAGIC score at Day 28 and remain a CR responder or PR responder on the total MAGIC score at Day 56.
  Total MAGIC staging for each of the 4 evaluable organs of skin, lower and upper GI tract, and liver ranges from 0 to 4, with higher number indicating a worse state of disease. (For complete staging criteria, see: Harris AC, et al. Biol Blood Marrow Transplant. 2016;22(1):4-10.)
Time Frame: Day 28 to Day 56
Population: Full Analysis Set: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants
  Lower GI MAGIC Score | 53.3 [26.6 to 78.7] | 33.3 [11.8 to 61.6] | 100 [2.5 to 100]
  Total MAGIC Score | 53.3 [26.6 to 78.7] | 33.3 [11.8 to 61.6] | 100 [2.5 to 100]

14. Secondary Outcome: Duration of Response From Day 56 on the Total MAGIC Score
Description: Duration of response from Day 56 on the total MAGIC score: defined as the interval from the Day 56 response (PR and CR; see definitions descriptions in Outcome Measure 12) to death or new systemic therapy for aGVHD (including an increase in steroids >2 mg/kg/day methylprednisolone [MP] equivalent), whichever occurs first, with at least 182 days of follow-up.
  Total MAGIC staging for each of the 4 evaluable organs of skin, lower and upper GI tract, and liver range from 0 to 4, with higher number indicating a worse state of disease. (For complete staging criteria, see: Harris AC, et al. Biol Blood Marrow Transplant. 2016;22(1):4-10.)
  Full range dates are censored. Censored = participants alive and without missing overall response assessment, initiation of additional systemic therapy for aGVHD or increase of >2 mg/kg/day MP equivalent in steroids. Subjects are right censored at their last follow-up visit.
Time Frame: From Day 56 up to 2 years of follow up after the first dose
Population: Full Analysis Set: all enrolled participants. Participants with a best response of CR or PR on the Total MAGIC Score from Day 56.
Measure: Median (Full Range); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 8 | 7 | 1
days | 483.0 [37 to 686] | NA [32 to 666] — Not estimable due to low number of events. | 64.0 [64 to 64]

15. Secondary Outcome: Duration of Response From Day 28 on the Total MAGIC Score
Description: Duration of response from Day 28 on the total MAGIC score: defined as the interval from the Day 28 response (PR and CR; see definitions descriptions in Outcome Measure 12) to death or new systemic therapy for aGVHD (including an increase in steroids >2 mg/kg/day methylprednisolone [MP] equivalent), whichever occurs first, with at least 182 days of follow-up.
  Total MAGIC staging for each of the 4 evaluable organs of skin, lower and upper GI tract, and liver range from 0 to 4, with higher number indicating a worse state of disease. (For complete staging criteria, see: Harris AC, et al. Biol Blood Marrow Transplant. 2016;22(1):4-10.) Full range dates are censored. Censored = participants alive and without missing overall response assessment, initiation of additional systemic therapy for aGVHD or increase of >2 mg/kg/day MP equivalent in steroids. Subjects are right censored at their last follow-up visit.
Time Frame: From Day 28 up to 2 years of follow up after the first dose
Population: Full Analysis Set: all enrolled participants. Participants with best response of CR or PR on the Total MAGIC Score from Day 28.
Measure: Median (Full Range); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 10 | 7 | 1
days | 511.0 [13 to 714] | NA [12 to 694] — Not estimable due to the low number of events. | 92.0 [92 to 92]

16. Secondary Outcome: Duration of Lower GI Response Per MAGIC Score
Description: Individual duration of lower GI response (either CR responder or PR responder, see Outcome Measure 10 description for details) counted from the first response to return to baseline or worse.
  Duration of lower GI response is defined as the duration from the first date a participant is identified as a Lower GI MAGIC Score CR or PR responder until the next date a subject is Lower GI MAGIC Score stable disease/progressed disease (SD/PD; i.e., return to baseline or worsening), experiences treatment failure, or dies, whichever occurs first.
Time Frame: Up to Day 147
Population: Full Analysis Set: all enrolled participants. Participants with best response of CR or PR on the Lower GI MAGIC Score.
Measure: Median (Full Range); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 13 | 13 | 1
days | 58.0 [1 to 729] | 22.0 [1 to 358] | 113.0 [113 to 113]

17. Secondary Outcome: Duration of Lower GI Response Per MAGIC Score In Retreated Participants
Description: Individual duration of lower GI response (either CR responder or PR responder, see Outcome Measure 10 description for details) counted from the first response to return to baseline or worse in participants that were re-treated with apraglutide because of a lower GI-aGVHD flare, counted from the first response after apraglutide restart to return to baseline or worse.
  Duration of lower GI response is defined as the duration from the first date a participant is identified as a Lower GI MAGIC Score CR or PR responder until the next date a subject is Lower GI MAGIC Score stable disease/progressed disease (SD/PD; i.e., return to baseline or worsening), experiences treatment failure, or dies, whichever occurs first.
Time Frame: Up to Day 147
Population: Full Analysis Set: all enrolled participants. Participants who were re-treated with apraglutide because of a lower GI-aGVHD flare.
Measure: Number; unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 0 | 0 | 1
days |  |  | NA — Participant was re-treated but did not respond, therefore a duration of response for retreated participants could not be calculated.

18. Secondary Outcome: Time to Partial or Complete Lower GI Response (PR or CR) Per MAGIC Score
Description: Lower GI (Stool Output/Day) MAGIC Stages are 0: <500 mL/day or <3/episodes/day; 1: 500-999 mL/day or 3-4/episodes/day; 2: 1000-1500 mL/day or 5-7/episodes/day; 3: >1500 mL/day or >7/episodes/day; 4: Severe abdominal pain with or without ileus or grossly bloody stool (regardless of volume).
  CR: Score of 0 in lower GI tract MAGIC stage that indicates complete resolution of all signs and symptoms of aGVHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGVHD. PR: Improvement of one stage in lower GI tract MAGIC stage without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response, or non-response of aGVHD.
Time Frame: From first injection of apraglutide up to Day 57
Population: Full Analysis Set: all enrolled participants. Participants with a complete and/or partial lower GI response per MAGIC Score.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 13 | 13 | 1
days
  Time to Complete or Partial Lower GI Response | 14.2 (8.33) | 16.6 (10.60) | 9.0 (NA) — Only 1 participant in this arm.
  Time to Partial Lower GI Response: number analyzed (Participants) | 10 | 11 | 0
  Time to Partial Lower GI Response | 14.0 (7.72) | 22.9 (15.64) |
  Time to Complete Lower GI Response: number analyzed (Participants) | 10 | 8 | 1
  Time to Complete Lower GI Response | 41.9 (31.24) | 23.8 (18.61) | 9.0 (NA) — Only 1 participant in this arm.

19. Secondary Outcome: Best Overall Lower GI Response and Total Response at Any Time Point Up to and Including Day 91
Description: Overall response rate on the Lower GI MAGIC Score is defined as the percentage of participants who had a response (either CR responder or PR responder, see Outcome Measure 10 description for details) on the lower GI score. Overall response rate on the Total MAGIC Score is defined as the percentage of participants who had a response (either CR responder or PR responder, see Outcome Measure 12 description for details) on the total MAGIC score. Best overall lower GI response and total response is defined as overall response (PR or CR) at any time point up to and including Day 91 and before the start of additional systemic therapy for lower GI aGVHD.
  MAGIC staging for each of the 4 evaluable organs of skin, lower and upper GI tract, and liver ranges from 0 to 4, with higher number indicating a worse state of disease. (For complete staging criteria, see: Harris AC, et al. Biol Blood Marrow Transplant. 2016;22(1):4-10.)
Time Frame: From first injection of apraglutide up to Day 91
Population: Full Analysis Set: All enrolled participants with a response and an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 13 | 13 | 1
percentage of participants
  Best Overall Lower GI Response = CR | 66.7 [38.4 to 88.2] | 53.3 [26.6 to 78.7] | 100 [2.5 to 100]
  Best Overall Lower GI Response = PR | 20.0 [4.3 to 48.1] | 33.3 [11.8 to 61.6] | 0 [0 to 97.5]
  Best Overall Response per Total MAGIC Score = CR | 60.0 [32.3 to 83.7] | 53.3 [26.6 to 78.7] | 100 [2.5 to 100]
  Best Overall Response per Total MAGIC Score = PR | 33.3 [11.8 to 61.6] | 40.0 [16.3 to 67.7] | 0 [0 to 97.5]

20. Secondary Outcome: Failure-Free Survival Post-First Dose of Apraglutide
Description: Failure free survival is defined as time from first dose until death, hematologic malignancy relapse/progression, or treatment failure, whichever comes first. Treatment failure is reported when additional systemic therapies are used for any earlier progression, mixed response or stable aGVHD.
Time Frame: Baseline up to 2 years
Population: Full Analysis Set: all enrolled participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
days | 539.0 [97.0 to NA] — Not estimable due to the low number of events. | 103.0 [45.0 to NA] — Not estimable due to the low number of events. | 121.0 [NA to NA] — Only one participant in this arm.

21. Secondary Outcome: Time to Non-Relapse Mortality up to 2 Years Post Treatment Start
Description: Non-relapse mortality is defined as time from first dose until death without preceding hematologic relapse.
Time Frame: From first dose of apraglutide up to 2 years
Population: Full Analysis Set: all enrolled participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
days | NA [539.0 to NA] — Not estimable due to the low number of events. | NA [103.0 to NA] — Not estimable due to the low number of events. | 175.0 [NA to NA] — Only 1 participant in this arm.

22. Secondary Outcome: Overall Survival
Description: Overall survival is calculated as the time from first dose of apgraglutide to death.
Time Frame: Baseline up to 2 years post-first dose of apraglutide
Population: Full Analysis Set: all enrolled participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
days | NA [539.0 to NA] — Not estimable due to the low number of events. | 169.0 [45.0 to NA] — Not estimable due to the low number of events. | 175.0 [NA to NA] — Only 1 participant in this arm.

23. Secondary Outcome: Percentage of Participants With Hematologic Malignancy Relapse/Progression
Time Frame: Baseline to 2 years
Population: Full Analysis Set: all enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants | 6.7 | 6.7 | 0

24. Secondary Outcome: Percentage of Participants With Graft Failure Up to 2 Years Post-first Dose of Apraglutide
Description: Primary graft failure:
  Absolute neutrophil count < 0.5 × 10^9/L by Day 28 Hemoglobin <80 g/L and platelets < 20 × 10^9/L Reduced intensity conditioning: Confirmation of donor cell origin is required Cord blood transplant: Up to Day +42
  Secondary graft failure:
  Absolute neutrophil count < 0.5 × 10^9/L after initial engraftment not related to relapse, infection, or drug toxicity Reduced intensity conditioning: Loss of donor hematopoiesis to < 5%
Time Frame: From first dose of apraglutide up to 2 years post-first dose
Population: Full Analysis Set: all enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants | 0 | 6.7 | 0

25. Secondary Outcome: Percentage of Participants Who Experienced Lower-GI Flare by Day 182 After Earlier Cessation of Treatment Due to CR
Description: Incidence of lower GI-aGVHD flare up to Day 182 after the first apraglutide dose following earlier cessation due to complete lower GI-aGVHD response. A lower GI-aGVHD flare is defined as any increase in signs or symptoms of lower GI-aGVHD that is sustained for >24 hours after apraglutide treatment completion following a CR or PR in the lower GI (see Outcome Measure 10 description for details) and requires re-escalation of immunosuppressive therapy (e.g., corticosteroid, calcineurin inhibitors and/or ruxolitinib dosing).
Time Frame: From first apraglutide dose up to Day 182
Population: Full Analysis Set: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apraglutide Low Dose: Low-dose, weight-based apraglutide SC injections (1.4 to 2.5 mg) once weekly for up to 13 weeks (with optional treatment up to an additional 13 weeks), for participants with body weight of more than 50.0 kg.
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
percentage of participants | 0 [0 to 21.8] | 0 [0 to 21.8] | 100 [2.5 to 100]

26. Secondary Outcome: Cumulative Ruxolitinib (RUX) and Systemic Steroid (SS) Doses From Start of the RUX Treatment up to Day 91 After the First Dose of Apraglutide
Description: Concomitant treatment with any systemic GVHD therapy other than SS and RUX was prohibited. The exact dose of SS and RUX taken throughout the trial was recorded in the case report form, including any dose adjustments. Systemic steroid dose was computed using the converted systemic methylprednisolone equivalent dose.
Time Frame: From start of the RUX treatment up to Day 91 after the first dose of apraglutide
Population: Safety Analysis Set: All the randomized participants exposed to at least 1 dose of apraglutide.Participant with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
mg/kg
  RUX : Baseline - Day 7 | 1.724 (0.6375) | 1.580 (0.4490) | 1.935 (NA) — Only 1 participant in this arm.
  RUX : Day 7 - Day 14 | 1.714 (0.5747) | 1.369 (0.6378) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 14 - Day 21: number analyzed (Participants) | 15 | 14 | 1
  RUX : Day 14 - Day 21 | 1.444 (0.8280) | 1.212 (0.7907) | 2.796 (NA) — Only 1 participant in this arm.
  RUX : Day 21 - Day 28: number analyzed (Participants) | 14 | 14 | 1
  RUX : Day 21 - Day 28 | 1.549 (0.8357) | 1.020 (0.8496) | 3.011 (NA) — Only 1 participant in this arm.
  RUX : Day 28 - Day 35: number analyzed (Participants) | 14 | 13 | 1
  RUX : Day 28 - Day 35 | 1.523 (0.8421) | 0.911 (0.8010) | 2.581 (NA) — Only 1 participant in this arm.
  RUX : Day 35 - Day 42: number analyzed (Participants) | 14 | 11 | 1
  RUX : Day 35 - Day 42 | 1.355 (0.9044) | 0.927 (0.9531) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 42 - Day 49: number analyzed (Participants) | 13 | 10 | 1
  RUX : Day 42 - Day 49 | 1.357 (0.9557) | 1.062 (0.8769) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 49 - Day 56: number analyzed (Participants) | 11 | 10 | 1
  RUX : Day 49 - Day 56 | 1.308 (0.9458) | 1.038 (0.8778) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 56 - Day 63: number analyzed (Participants) | 10 | 10 | 1
  RUX : Day 56 - Day 63 | 1.185 (0.8464) | 1.049 (0.9070) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 63 - Day 70: number analyzed (Participants) | 9 | 9 | 1
  RUX : Day 63 - Day 70 | 1.204 (0.9220) | 1.114 (0.8958) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 70 - Day 77: number analyzed (Participants) | 9 | 9 | 1
  RUX : Day 70 - Day 77 | 1.169 (0.7941) | 1.114 (0.8958) | 1.505 (NA) — Only 1 participant in this arm.
  RUX : Day 77 - Day 84: number analyzed (Participants) | 9 | 9 | 1
  RUX : Day 77 - Day 84 | 1.162 (0.7507) | 1.033 (0.7451) | 0.968 (NA) — Only 1 participant in this arm.
  RUX : Day 84 - Day 91: number analyzed (Participants) | 8 | 9 | 1
  RUX : Day 84 - Day 91 | 1.247 (0.7381) | 1.049 (0.7397) | 1.505 (NA) — Only 1 participant in this arm.
  SS : Baseline - Day 7 | 7.951 (4.6608) | 9.482 (4.2267) | 15.484 (NA) — Only 1 participant in this arm.
  SS : Day 7 - Day 14 | 5.931 (4.5259) | 5.543 (3.9627) | 13.118 (NA) — Only 1 participant in this arm.
  SS : Day 14 - Day 21: number analyzed (Participants) | 15 | 14 | 1
  SS : Day 14 - Day 21 | 4.924 (3.9327) | 3.938 (2.6529) | 11.398 (NA) — Only 1 participant in this arm.
  SS : Day 21 - Day 28: number analyzed (Participants) | 15 | 14 | 1
  SS : Day 21 - Day 28 | 3.661 (3.3871) | 2.864 (2.4736) | 9.032 (NA) — Only 1 participant in this arm.
  SS : Day 28 - Day 35: number analyzed (Participants) | 14 | 12 | 1
  SS : Day 28 - Day 35 | 3.066 (2.9184) | 2.057 (1.4276) | 9.892 (NA) — Only 1 participant in this arm.
  SS : Day 35 - Day 42: number analyzed (Participants) | 14 | 11 | 1
  SS : Day 35 - Day 42 | 2.675 (2.7542) | 1.687 (1.6041) | 8.430 (NA) — Only 1 participant in this arm.
  SS : Day 42 - Day 49: number analyzed (Participants) | 13 | 10 | 1
  SS : Day 42 - Day 49 | 2.124 (2.2079) | 1.026 (0.8366) | 6.366 (NA) — Only 1 participant in this arm.
  SS : Day 49 - Day 56: number analyzed (Participants) | 11 | 10 | 1
  SS : Day 49 - Day 56 | 1.681 (2.1940) | 0.882 (0.6197) | 6.022 (NA) — Only 1 participant in this arm.
  SS : Day 56 - Day 63 | 1.586 (1.1506) | 0.988 (0.5212) | 5.849 (NA) — Only 1 participant in this arm.
  SS : Day 63 - Day 70: number analyzed (Participants) | 7 | 8 | 1
  SS : Day 63 - Day 70 | 1.069 (0.8051) | 0.988 (0.8091) | 5.419 (NA) — Only 1 participant in this arm.
  SS : Day 70 - Day 77: number analyzed (Participants) | 7 | 8 | 1
  SS : Day 70 - Day 77 | 1.802 (2.1332) | 0.800 (0.7199) | 5.419 (NA) — Only 1 participant in this arm.
  SS : Day 77 - Day 84: number analyzed (Participants) | 7 | 6 | 1
  SS : Day 77 - Day 84 | 1.422 (2.0178) | 0.945 (0.7223) | 6.882 (NA) — Only 1 participant in this arm.
  SS : Day 84 - Day 91: number analyzed (Participants) | 6 | 6 | 1
  SS : Day 84 - Day 91 | 1.353 (1.8912) | 1.021 (0.6495) | 8.430 (NA) — Only 1 participant in this arm.

27. Secondary Outcome: Number of Participants With Treatment-Emergent Infections and Sepsis
Time Frame: From baseline to Day 91 and overall (up to 2 years after the first dose of apraglutide)
Population: Safety Analysis Set: All the randomized participants exposed to at least 1 dose of apraglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
Number analyzed (Participants) | 15 | 15 | 1
Participants
  Between Baseline and Day 91 : Infections | 8 | 14 | 1
  Between Baseline and Day 91 : Sepsis | 3 | 2 | 0
  Between Baseline and Study End : Infections | 8 | 15 | 1
  Between Baseline and Study End : Sepsis | 3 | 3 | 0

ADVERSE EVENTS:
Time Frame: Screening (up to 12 weeks) through End of Trial (up to 2 years/104 weeks) for a total of up to 116 weeks
Arm/Group | Apraglutide Low Dose | Apraglutide High Dose | Apraglutide Standard Dose
All-Cause Mortality (participants affected / at risk) | 3/15 | 6/15 | 1/1
Serious Adverse Events (participants affected / at risk) | 6/15 | 15/15 | 1/1
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apraglutide Low Dose (N=15) | Apraglutide High Dose (N=15) | Apraglutide Standard Dose (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Bacteroides bacteraemia (Infections and infestations) | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 0 | 1 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Air embolism (Vascular disorders) | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apraglutide Low Dose (N=15) | Apraglutide High Dose (N=15) | Apraglutide Standard Dose (N=1)
Anaemia (Blood and lymphatic system disorders) | 6 | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 7 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 4 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 3 | 1
Epstein-Barr virus infection reactivation (Infections and infestations) | 3 | 3 | 0
Oral candidiasis (Infections and infestations) | 1 | 3 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0
COVID-19 (Infections and infestations) | 0 | 3 | 0
Cystitis viral (Infections and infestations) | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
BK virus infection (Infections and infestations) | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 1 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Oesophageal infection (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Polyomavirus viraemia (Infections and infestations) | 0 | 1 | 0
Pyuria (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis bacterial (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis mycoplasmal (Infections and infestations) | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 0 | 1
Oedema peripheral (General disorders) | 7 | 10 | 0
Fatigue (General disorders) | 4 | 2 | 0
Pyrexia (General disorders) | 3 | 0 | 1
Asthenia (General disorders) | 0 | 2 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 0
Ileus (Gastrointestinal disorders) | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal wall oedema (Gastrointestinal disorders) | 1 | 0 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Oral blood blister (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 1 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 2 | 1
Blood creatinine increased (Investigations) | 2 | 2 | 0
Lipase increased (Investigations) | 3 | 1 | 0
Amylase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 2 | 0
Transaminases increased (Investigations) | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
BK polyomavirus test positive (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 1 | 0
Candida test positive (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Pseudomonas test positive (Investigations) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 2 | 1
Graft versus host disease oral (Immune system disorders) | 1 | 2 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Depression (Psychiatric disorders) | 3 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 3 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Dysphemia (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 3 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Perineal fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vulva cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The administered doses during the study were lower than protocol specified doses. This difference was due to dilution effects and injection-related volume loss during injection preparation, and were applied consistently across all injections and participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT05415410/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05415410/SAP_001.pdf